CLINICAL TRIAL: NCT01909453
Title: A 2-part Phase III Randomized, Open Label, Multicenter Study of LGX818 Plus MEK162 Versus Vemurafenib and LGX818 Monotherapy in Patients With Unresectable or Metastatic BRAF V600 Mutant Melanoma
Brief Title: Study Comparing Combination of LGX818 Plus MEK162 Versus Vemurafenib and LGX818 Monotherapy in BRAF Mutant Melanoma
Acronym: COLUMBUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMEK162B2301; C4221004 (Other: Alias Study Number); 2013-001176-38 (EudraCT Number)
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Results first posted 2021-07-12 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Melanoma
Keywords: Melanoma; Cutaneous melanoma; Skin disease; Skin cancer; Skin Neoplasms; Neoplasm Metastasis; BRAF mutant; BRAF V600E; BRAF V600K; Cancer; LGX818; MEK162; vemurafenib; combination; BRAF inhibitor; resistance; The combination of a selective BRAF- and a MEK1/2-inhibitor; Prior immunotherapy; MEK inhibitor; Phase III; Combo 300, Combo 450
MeSH Terms: conditions — Melanoma; Skin Diseases; Skin Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — encorafenib; binimetinib; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- LGX818 450 mg + MEK162 (Experimental): LGX818 450 mg QD + MEK162 45 mg BID
  Interventions: Drug: LGX818; Drug: MEK162
- Vemurafenib (Active Comparator): Vemurafenib 960 mg BID
  Interventions: Drug: vemurafenib
- LGX818 300 mg + MEK162 (Experimental): LGX818 300 mg QD + MEK162 45 mg BID
  Interventions: Drug: LGX818; Drug: MEK162
- LGX818 (Experimental): LGX818 300 mg QD
  Interventions: Drug: LGX818

INTERVENTIONS:
Drug: LGX818 — LGX818- Orally 100 mg and 50 mg capsules
  Arms: LGX818; LGX818 300 mg + MEK162; LGX818 450 mg + MEK162
Drug: MEK162 — MEK162- Orally 15 mg tablets
  Arms: LGX818 300 mg + MEK162; LGX818 450 mg + MEK162
Drug: vemurafenib — Tablets in bottles or blisters 240 mg
  Other Names: Zelboraf; PLX4032; RO5185426
  Arms: Vemurafenib

SUMMARY:
This is 2-part, randomized, open label, multi-center, parallel group, phase III study comparing the efficacy and safety of LGX818 plus MEK162 to vemurafenib and LGX818 monotherapy in patients with locally advanced unresectable or metastatic melanoma with BRAF V600 mutation. A total of approximately 900 patients will be randomized.

Part 1:

Patients will be randomized in a 1:1:1 ratio to one of 3 treatment arms:

1. LGX818 450 mg QD plus MEK162 45 mg BID (denoted as Combo 450 arm)
2. LGX818 300 mg QD monotherapy (denoted as LGX818 arm) or
3. vemurafenib 960 mg BID (denoted as vemurafenib arm)

Part 2:

Patients will be randomized in a 3:1 ratio to one of the 2 treatment arms:

1. LGX818 300 mg QD plus MEK162 45 mg BID (denoted as Combo 300 arm) or
2. LGX818 300 mg QD monotherapy (denoted as LGX818 arm)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced, unresectable or metastatic cutaneous melanoma or unknown primary melanoma (AJCC Stage IIIB, IIIC, or IV)
* Presence of BRAF V600E or V600K mutation in tumor tissue prior to randomization
* Naïve untreated patients or patients who have progressed on or after prior first line immunotherapy for resectable locally advanced or metastatic melanoma; prior adjuvant therapy is permitted (e.g. IFN, IL-2 therapy, any other immunotherapy, radiotherapy or chemotherapy), except the administration of BRAF or MEK inhibitors
* Evidence of at least one measurable lesion as detected by radiological or photographic methods
* ECOG performance status of 0 or 1
* Adequate bone marrow, organ function, cardiac and laboratory parameters
* Normal functioning of daily living activities

Exclusion Criteria:

* Any untreated central nervous system (CNS) lesion
* Uveal and mucosal melanoma
* History of leptomeningeal metastases
* History of or current evidence of central serous retinopathy (CSR), retinal vein occlusion (RVO) or history of retinal degenerative disease
* Any previous systemic chemotherapy treatment, extensive radiotherapy or investigational agent other than immunotherapy, or patients who have received more than one line of immunotherapy for locally advanced unresectable or metastatic melanoma; Ipilimumab (adjuvant) or other immunotherapy treatment must have ended at least 6 weeks prior to randomization
* History of Gilbert's syndrome
* Prior therapy with a BRAF inhibitor and/or a MEK- inhibitor
* Impaired cardiovascular function or clinically significant cardiovascular diseases
* Uncontrolled arterial hypertension despite medical treatment
* HIV positive or active Hepatitis B, and/or active Hepatitis C
* Impairment of gastrointestinal function
* Patients with neuromuscular disorders that are associated with elevated CK
* Pregnant or nursing (lactating) women
* Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 921 (Actual)
Dates: Start 2013-09-12 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2024-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (280):
- United States (49):
  - Retinal Consultants of Alabama P.C., Birmingham, Alabama
  - UAB Callahan Eye Hospital, Birmingham, Alabama
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - UAB The Kirklin Clinic, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Oncology Associates, Tucson, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Highlands Oncology Group - Fayetteville, Springdale, Arkansas
  - UC Irvine Medical Center, Orange, California
  - Rocky Mountain Cancer Centers (Williams) - USOR, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers (Williams) - USOR, Denver, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Specialty Eye Care, Parker, Colorado
  - Rocky Mountain Cancer Centers, Pueblo, Colorado
  - University Cancer Institute, Boynton Beach, Florida
  - University of Miami, Miami, Florida
  - Eye & Ear Infirmary- Opthalmology, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System - Investigational Drug Service, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - University of Illinois Medical Center, Chicago, Illinois
  - Oncology Specialists, SC, Niles, Illinois
  - Goshen Center For Cancer Care, Goshen, Indiana
  - Lack's Cancer Center at Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Mercy Health Hauenstein Neuroscience Center Neuro-Ophthalmology (Clinic), Grand Rapids, Michigan
  - Retina Specialists of Michigan, Grand Rapids, Michigan
  - Hattiesburg Clinic Oncology Hem, Hattiesburg, Mississippi
  - Jackson Oncology Associates - St. Dominic Hospital, Jackson, Mississippi
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Investigational Drug Service, Department of Pharmacy (Investigational Product), Rochester, New York
  - University of Rochester Medical Center - PPDS, Rochester, New York
  - Tulsa Cancer Institute PLLC, Tulsa, Oklahoma
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Sanford Cancer Center Oncology Clinic & Pharmacy, Sioux Falls, South Dakota
  - University of Tennessee Medical Center Cancer Institute, Knoxville, Tennessee
  - Dr. Dennis B. Kay (Ophthalmologist), Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Virginia Cancer Specialists, PC, Alexandria, Virginia
  - Virginia Cancer Specialists, Arlington, Virginia
  - Virginia Cancer Specialists (Leesburg) - USOR, Fairfax, Virginia
  - Northern Virginia Ophthalmology Associates, Falls Church, Virginia
  - Virginia Cancer Specialists, PC, Gainesville, Virginia
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
- Argentina (3):
  - Fundación CENIT para la Investigación en Neurociencias, CABA, Buenos Aires
  - Fundación Investigar, Buenos Aires, Ciudad Autónoma de Buenosaires
  - Instituto Médico Especializado Alexander Fleming, Buenos Aires, Ciudad Autónoma de Buenosaires
- Australia (6):
  - Lake Macquarie Private Hospital, Gateshead, New South Wales
  - Tasman Oncology Research, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - The Alfred Hospital, Prahran, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Brazil (8):
  - AMO - Assistência Multidisciplinar em Oncologia, Salvador, Estado de Bahia
  - Instituto de Medicina Integral Professor Fernando Figueira, Recife, Pernambuco
  - Associação Hospital de Caridade Ijuí, Ijuí, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre (HCPA) - PPDS, Porto Alegre, Rio Grande do Sul
  - Fundação PIO XII, Barretos, São Paulo
  - Liga Norte Riograndense Contra O Cancer, Natal
  - INCA Instituto Nacional de Cancer, Rio de Janeiro
  - Hospital BP Mirante, São Paulo
- Canada (8):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - SunnyBrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier De L'Universite De Montreal Hospital Notre Dame, Montreal, Quebec
  - CHUM Notrea Dame Hospital, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University Health center, Montreal, Quebec
  - CHU de Quebec-Universite Laval - L' Hotel - Dieu de Quebec, Québec
- Hospital Universitario San Ignacio, Bogotá, Bogota D.C., Colombia
- Czechia (5):
  - Fakultni nemocnice Ostrava, Ostrava, Moravskoslezský kraj
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Praha, Hlavní Mesto
  - Mou/Mmci - Ppds, Brno, South Moravian
  - Fakultni nemocnice Olomouc, Olomouc
  - General Faculty Hospital, Prague
- France (15):
  - CHU de Grenoble, Grenoble, Isère
  - CHRU de Lille - Hôpital Huriet, Lille, NORD
  - Centre Léon Bérard Centre Régional de Lutte Contre Le Cancer Rhône Alpes, Lyon, Rhone
  - Centre Hospitalier Le Mans, Le Mans, Sarthe
  - Institut Gustave Roussy, Villejuif, Val-de-marne
  - Hopital Saint Andre Unite de Cancerologie Service de Dermatologie, Bordeaux
  - Centre Hospitalier Universitaire Ambroise Paré, Boulogne-Billancourt
  - Groupe Hospitalier Archet I Et II, Nice
  - Hopital Lariboisiere, Paris
  - Institut Mutualiste Montsouris, Paris
  - Ophtalmologist office, Paris
  - Hôpital Saint louis, Paris
  - Hospices Civils de Lyon - Hopital Lyon Sud, Pierre-Bénite
  - CHU de Reims - Hôpital Robert Debré, Reims
  - Nouvel Hopital Civil, Strasbourg
- Germany (47):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - University Clinic Heidelberg - PPDS, Heidelberg, Baden-Wurttemberg
  - Klinikum Mannheim Universitätsklinikum gGmbH, Mannheim, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum Bayreuth GmbH, Bayreuth, Bavaria
  - LMU Klinikum, München, Bavaria
  - Hautklinik, Klinikum Nürnberg, Universitätsklinik der Paracelsus Medizinischen Privatuniversität, Nuremberg, Bavaria
  - Institut für Röntgendiagnostik, Regensburg, Bavaria
  - University Clinic Regensburg - PPDS, Regensburg, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Klinikum Kassel, Kassel, Hesse
  - Augenarztzentrum Buxtehude, Buxtehude, Lower Saxony
  - Elben Klinken Stade ? Buxtehude, Buxtehude, Lower Saxony
  - Augenklinik Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Institut für Diagnostische Radiologie, Neuroradiologie und Nuklearmedizin, Minden, North Rhine-Westphalia
  - Mühlenkreiskliniken - Johannes Wesling Klinikum Minden, Minden, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitatsklinikum Leipzig AoR, Leipzig, Saxony
  - Universitätsklinikum Magdeburg A.ö.R., Magdeburg, Saxony-Anhalt
  - Universitatsklinikum Schleswig-Holstein, Campus Lubeck, Lübeck, Schleswig-Holstein
  - Charite-Universitaetsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - University Hospital Carl Gustav Carus at the Technical University of Dresden, Dresden
  - Überörtliche Radiologische Gemeinschaftspraxis Dresden, Dresden
  - Klinik fur Hautkrankheiten und Allergologie, Helios Hauttumorzentrum Erfurt, Helios Klinikum Erfurt, Erfurt
  - Universitätsklinikum Essen, Essen
  - Goethe-University Frankfurt/Main, Frankfurt am Main
  - Universitätsklinikum Freiburg, Klinik für Radiologie, Freiburg im Breisgau
  - Institut für Diagnostische und Interventionelle Radiologie, Gera
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Klinik für Augenheilkunde, Gera
  - Universitätsklinik Hamburg Eppendorf, Hamburg
  - Augenärzte am Kröpcke, Hanover
  - Medizinische Hochschule Hannover (Hannover Medical School), Hanover
  - Institut für Diagnostische und Interventionelle Radilogie, Hanover
  - University Clinic Heidelberg - PPDS, Heidelberg
  - Universität des Saarlandes, Homburg
  - University Hospital Schleswig-Holstein, Campus Kiel, Kiel
  - Augenklinik Universitätsklinikum Mannheim, Mannheim
  - Augen-Praxis_Minden, Minden
  - Fachklinik Hornheide Abteilung für Internistische Onkologie und Hämatologie, Münster
  - Klinikum Nürnberg - Campus Nord, Nuremberg
  - Klinik & Poliklinik für Augenheilkunde, Regensburg
  - Universitätsklinikum Tübingen, Tübingen
  - Internistische Schwerpunktpraxis Kardiologie Hämatologie Onkologie, Ulm
  - Universitätsklinikum Ulm, Ulm
- Greece (2):
  - Laiko General Hospital of Athens, Athens
  - Metropolitan Hospital, Neo Faliro
- Hungary (4):
  - Debreceni Egyetem Klinikai Kozpont, Debrecen, Hajdú-Bihar
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
- Israel (3):
  - Sheba Medical Center - PPDS, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center - PPDS, Jerusalem
- Italy (27):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona-Umberto I G.M. Lancisi G. Salesi, Torrette Site, Ancona
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - Azienda Ospedaliero Universitaria Di Bologna Policlinico S Orsola Malpighi, Bologna, Emilia-Romagna
  - Policlinico Universitario Campus Biomedico Di Roma, Rome, Lazio
  - Istituto Nazionale Tumori Regina Elena, Rome, Lazio
  - Istituto Dermopatico dell'Immacolata IRCCS, Rome, Lazio
  - ASST degli Spedali Civili di Brescia - Spedali Civili di Brescia - INCIPIT - PIN, Brescia, Lombardy
  - Azienda Ospedaliera Ospedale Di Lecco, Lecco, Lombardy
  - Istituto Nazionale Dei Tumori, Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda, Milan, Lombardy
  - Azienda Ospedaliera San Gerardo, Monza, Lombardy
  - Fondazione del Piemonte per l'Oncologia (IRCCS), Candiolo, Torino
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Azienda Ospedaliera S Maria Di Terni, Terni, Umbria
  - Clinica Oculistica, Padua, Veneto
  - IRCCS Giovanni Paolo II Cancer Institute, Bari
  - ASST Papa Giovanni XXIII - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - IRCCS Az. Osp. Universitaria San Martino- IST, Genoa
  - Istituto Europeo Di Oncologia, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Giovanni Pascale, Napoli
  - Istituto Oncologico Veneto - I.R.C.C.S., Padua
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
  - Azienda Ospedaliera Civile Maria Paternò Arezzo Ragusa, Ragusa
  - S. C. Oncologia Medica Presidio Ospedaliero Maria Paterno Arezzo, Ragusa
  - Policlinico Universitario Campus Biomedico, Rome
  - Azienza Ospedaliera Universitaria Senese, Siena
  - Azienda Sanitaria Universitaria Integrata di Udine - PO Universitario Santa Maria della Misericordia, Udine
- Japan (5):
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Shinshu University Hospital, Matsumoto, Nagano
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - National Hospital Organization Osaka National Hospital, Osaka, Ôsaka
- Mexico (4):
  - Instituto Nacional de Cancerologia, Mexico City, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Cancun Oncology Center Galenia, Cancún, Quintana Roo
  - Medica Sur, S. A. B de C. V. (Centro de Investigación Farmacológica y Biotecnológica CIF-BIOTEC), México
- Netherlands (15):
  - Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland
  - Amphia Ziekenhuis, Breda, North Brabant
  - Maxima Medisch Centrum, Eindhoven, North Brabant
  - VU Medisch Centrum, Amsterdam, North Holland
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Isala Zwolle, Zwolle, Overijssel
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Medisch Spectrum Twente - Hospital, Ariënsplein Enschede
  - Medisch Spectrum Twente, Enschede
  - Universitair Medisch Centrum Groningen, Groningen
  - Zuyderland Medisch Centrum - Heerlen, Heerlen
  - Leids Universitair Medisch Centrum, Leiden
  - Maastricht University Medical Center, Maastricht
  - Erasmus MC, Rotterdam
  - Erasmus MC-Daniel den Hoed Oncologisch Centrum, Rotterdam
- Norway (3):
  - Oslo universitetssykehus HF, Utprøvingsenheten, Oslo
  - Oslo universitetssykehus HF, Oslo
  - Oslo Myeloma Center - PPDS, Oslo
- Poland (3):
  - Centrum Medyczne MAVIT Sp. z o.o., Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie, Warsaw, Masovian Voivodeship
  - Lux Med, Warsaw
- Portugal (5):
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, E.P.E., Lisbon, Lisbon District
  - Hospital Garcia de Orta*E.P.E., Almada, Setúbal District
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe - PPDS, Lisbon
  - Centro Hospitalar de Lisboa Norte, E.P.E- Hospital de Santa Maria, Lisbon
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe - PPDS, Porto
- Russia (4):
  - Russian Oncology Research Center n a N N Blokhin, Moscow
  - Ryazan Clinical Hospital n.a. Semashko, Ryazan
  - Ryazan Regional Clinical Oncology Dispensary, Ryazan
  - Scientific Research Institute of Oncology n.a. N.N. Petrov, Saint Petersburg
- Singapore (4):
  - National Cancer Centre - 30 Hospital Blvd, Singapore
  - Singapore General Hospital (SGH), Singapore
  - National Cancer Centre Singapore, Singapore
  - Singapore National Eye Research Centre, Singapore
- Slovakia (2):
  - Narodny onkologicky ustav - PPDS, Bratislava
  - POKO POPRAD, s.r.o., Poprad
- South Africa (2):
  - Steve Biko Academic Hospital, Pretoria
  - Mary Potter Oncology Centre, Pretoria
- South Korea (4):
  - Samsung Medical Center - PPDS, Gangnam-gu, Seoul Teugbyeolsi
  - Asan Medical Center - PPDS, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
- Spain (27):
  - Hospital Universitario de Jerez, Jerez de la Frontera, Andalusia
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Cetir, Centre Mèdic, S.L, Barcelona, Catalonia
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Nuestra Señora de Valme, Seville, Sevilla
  - Hospital Universitario A Coruña, A Coruña
  - Hospital General Universitario Dr. Balmis, Alicante
  - Centro de Oftalmologia Barraquer, Barcelona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Onkologikoa, Donostia / San Sebastian
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Civil (Hospital Regional Universitario de Malaga), Málaga
  - Hospital Universitario Nuestra Sra de La Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Fundacion Instituto Valenciano de Oncologia, Valencia
- Sweden (6):
  - Gävle Sjukhus, Gävle
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Universitetssjukhuset i Linköping, Linköping
  - Skanes Universitetssjukhus Lund, Lund
  - Karolinska Universitetssjukhuset Solna, Solna
  - Uppsala Universitet, Uppsala
- Switzerland (2):
  - Inselspital Bern, Bern
  - Universitätsspital Zürich, Zurich Flughafen
- Turkey (Türkiye) (4):
  - Gazi University Medical Faculty Gazi Hospital, Ankara
  - Ege University Medical Faculty, Bornova
  - Ege University Medical aculty, Izmir
  - Sifa Universitesi Bornova Egitim Arastirma Hastanesi, Izmir
- United Kingdom (12):
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - The Royal Marsden NHS Foundation Trust, London, Chelsea
  - Mount Vernon Hospital, Northwood, London, CITY of
  - Royal Surrey County Hospital, Guildford, Surrey
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral
  - Weston Park Hospital, Sheffield, YORK
  - Broomfield Hospital, Broomfield
  - St James University Hospital, Leeds
  - Royal Free Hospital, London
  - The Christie NHS Foundation Trust - PPDS, Manchester
  - Churchill Hospital, Oxford
  - Royal Preston Hospital - NWCRN- PPDS, Preston

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Augustyn K, Joseph J, Patel AB, Razmandi A, Ali AN, Tawbi HA. Treatment experience with encorafenib plus binimetinib for BRAF V600-mutant metastatic melanoma: management insights for clinical practice. Melanoma Res. 2023 Oct 1;33(5):406-416. doi: 10.1097/CMR.0000000000000891. Epub 2023 Aug 3. PMID 37534686
- [Derived] Ascierto PA, Dummer R, Gogas HJ, Arance A, Mandala M, Liszkay G, Garbe C, Schadendorf D, Krajsova I, Gutzmer R, Chiarion-Sileni V, Dutriaux C, de Groot JWB, Yamazaki N, Loquai C, Robert C, Flaherty KT. Contribution of MEK Inhibition to BRAF/MEK Inhibitor Combination Treatment of BRAF-Mutant Melanoma: Part 2 of the Randomized, Open-Label, Phase III COLUMBUS Trial. J Clin Oncol. 2023 Oct 10;41(29):4621-4631. doi: 10.1200/JCO.22.02322. Epub 2023 Jul 28. PMID 37506329
- [Derived] Dummer R, Flaherty KT, Robert C, Arance A, B de Groot JW, Garbe C, Gogas HJ, Gutzmer R, Krajsova I, Liszkay G, Loquai C, Mandala M, Schadendorf D, Yamazaki N, Pietro AD, Cantey-Kiser J, Edwards M, Ascierto PA. COLUMBUS 5-year update: a randomized, open-label, phase III trial of encorafenib plus binimetinib versus vemurafenib or encorafenib in patients with BRAF. Future Oncol. 2023 May;19(16):1091-1098. doi: 10.2217/fon-2022-1258. Epub 2023 Jun 13. PMID 37309702
- [Derived] Li SN, Wan X, Peng LB, Li YM, Li JH. Cost-effectiveness of immune checkpoint inhibition and targeted treatment in combination as adjuvant treatment of patient with BRAF-mutant advanced melanoma. BMC Health Serv Res. 2023 Jan 18;23(1):49. doi: 10.1186/s12913-023-09058-7. PMID 36653848
- [Derived] Dummer R, Flaherty KT, Robert C, Arance A, de Groot JWB, Garbe C, Gogas HJ, Gutzmer R, Krajsova I, Liszkay G, Loquai C, Mandala M, Schadendorf D, Yamazaki N, di Pietro A, Cantey-Kiser J, Edwards M, Ascierto PA. COLUMBUS 5-Year Update: A Randomized, Open-Label, Phase III Trial of Encorafenib Plus Binimetinib Versus Vemurafenib or Encorafenib in Patients With BRAF V600-Mutant Melanoma. J Clin Oncol. 2022 Dec 20;40(36):4178-4188. doi: 10.1200/JCO.21.02659. Epub 2022 Jul 21. PMID 35862871
- [Derived] Gogas H, Dummer R, Ascierto PA, Arance A, Mandala M, Liszkay G, Garbe C, Schadendorf D, Krajsova I, Gutzmer R, Sileni VC, Dutriaux C, Yamazaki N, Loquai C, Queirolo P, Jan de Willem G, Sellier AT, Suissa J, Murris J, Gollerkeri A, Robert C, Flaherty KT. Quality of life in patients with BRAF-mutant melanoma receiving the combination encorafenib plus binimetinib: Results from a multicentre, open-label, randomised, phase III study (COLUMBUS). Eur J Cancer. 2021 Jul;152:116-128. doi: 10.1016/j.ejca.2021.04.028. Epub 2021 Jun 4. PMID 34091420
- [Derived] Gogas HJ, Flaherty KT, Dummer R, Ascierto PA, Arance A, Mandala M, Liszkay G, Garbe C, Schadendorf D, Krajsova I, Gutzmer R, Sileni VC, Dutriaux C, de Groot JWB, Yamazaki N, Loquai C, Gollerkeri A, Pickard MD, Robert C. Adverse events associated with encorafenib plus binimetinib in the COLUMBUS study: incidence, course and management. Eur J Cancer. 2019 Sep;119:97-106. doi: 10.1016/j.ejca.2019.07.016. Epub 2019 Aug 19. PMID 31437754
- [Derived] Dummer R, Ascierto PA, Gogas HJ, Arance A, Mandala M, Liszkay G, Garbe C, Schadendorf D, Krajsova I, Gutzmer R, Chiarion Sileni V, Dutriaux C, de Groot JWB, Yamazaki N, Loquai C, Moutouh-de Parseval LA, Pickard MD, Sandor V, Robert C, Flaherty KT. Overall survival in patients with BRAF-mutant melanoma receiving encorafenib plus binimetinib versus vemurafenib or encorafenib (COLUMBUS): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2018 Oct;19(10):1315-1327. doi: 10.1016/S1470-2045(18)30497-2. Epub 2018 Sep 12. PMID 30219628
- [Derived] Dummer R, Ascierto PA, Gogas HJ, Arance A, Mandala M, Liszkay G, Garbe C, Schadendorf D, Krajsova I, Gutzmer R, Chiarion-Sileni V, Dutriaux C, de Groot JWB, Yamazaki N, Loquai C, Moutouh-de Parseval LA, Pickard MD, Sandor V, Robert C, Flaherty KT. Encorafenib plus binimetinib versus vemurafenib or encorafenib in patients with BRAF-mutant melanoma (COLUMBUS): a multicentre, open-label, randomised phase 3 trial. Lancet Oncol. 2018 May;19(5):603-615. doi: 10.1016/S1470-2045(18)30142-6. Epub 2018 Mar 21. PMID 29573941

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: LGX818 450 mg QD+MEK162 45 mg BID (Combo 450): Participants received 450 milligram (mg) of LGX818 orally once daily (QD) along with 45 mg of MEK162 twice daily (BID) for each 28 day treatment cycle until progressive disease (PD) as confirmed by Blinded Independent Review Committee (BIRC), withdrawal of consent, intolerable toxicity, study discontinuation, lost to follow-up or death.
- Part 1: LGX818 300 mg; Part 2: LGX818 300 mg: Participants received 300 mg of LGX818 orally once daily for each 28 day treatment cycle until PD as confirmed by BIRC, withdrawal of consent, intolerable toxicity, study discontinuation, lost to follow-up or death.
- Part 1: Vemurafenib 960 mg BID: Participants received 960 mg of LGX818 according to the locally approved prescribing information twice daily for each 28 day treatment cycle until PD as confirmed by BIRC, withdrawal of consent, intolerable toxicity, study discontinuation, lost to follow-up or death.
- Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300): Participants received 300 mg of LGX818 orally once daily along with 45 mg of MEK162 twice daily for each 28 day treatment cycle until PD as confirmed by BIRC, withdrawal of consent, intolerable toxicity, study discontinuation, lost to follow-up or death.
Period: Overall Study
Arm/Group | Part 1: LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg
Started | 192 | 194 | 191 | 258 | 86
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 192 | 194 | 191 | 258 | 86
Not completed — Ongoing | 118 | 103 | 83 | 164 | 50
Not completed — Death | 69 | 74 | 88 | 86 | 29
Not completed — Lost to Follow-up | 3 | 4 | 4 | 3 | 3
Not completed — Withdrawal by Subject | 2 | 13 | 16 | 5 | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Total
Number analyzed (Participants) | 192 | 194 | 191 | 258 | 86 | 921
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 132 | 154 | 140 | 175 | 60 | 661
  >=65 years | 60 | 40 | 51 | 83 | 26 | 260
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 86 | 80 | 107 | 42 | 392
  Male | 115 | 108 | 111 | 151 | 44 | 529

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Progression Free Survival (PFS) by Blinded Independent Review Committee (BIRC) in Combo 450 Group as Compared to Vemurafenib Group
Description: PFS was defined as the time from the date of randomization to the date of the first documented disease progression (PD) or death due to any cause, whichever occurs first. PFS was determined based on tumor assessment (RECIST version 1.1 criteria) as per BIRC/central review and survival information. If a participant did not had an event at the time of the analysis cut-off or at the start of any new anti-cancer therapy, data was censored at the date of last adequate tumor assessment. PD was defined as at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must demonstrate an absolute increase of at least 5 square millimeter (mm^2).
Time Frame: From randomization until documented disease progression (PD), initiation of new anti-cancer therapy, censoring date or death, whichever occurred first (up to 29 months)
Population: FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450): Participants received 450 milligram (mg) of LGX818 orally once daily (QD) along with 45 mg of MEK162 twice daily (BID) for each 28 day treatment cycle until progressive disease (PD) as confirmed by Blinded Independent Review Committee (BIRC), withdrawal of consent, intolerable toxicity, study discontinuation, lost to follow-up or death.
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: Vemurafenib 960 mg BID
Number analyzed (Participants) | 192 | 191
months | 14.9 [11.0 to 18.5] | 7.3 [5.6 to 8.2]

2. Primary Outcome: Part 1: Progression Free Survival (PFS) by Blinded Independent Review Committee (BIRC) in Combo 450 Group as Compared to LGX818 Group
Description: PFS was defined as the time from the date of randomization to the date of the first documented disease progression (PD) or death due to any cause, whichever occurs first. PFS was determined based on tumor assessment (RECIST version 1.1 criteria) as per BIRC and survival information. If a participant did not had an event at the time of the analysis cut-off or at the start of any new anti-cancer therapy, data was censored at the date of last adequate tumor assessment. PD was defined as at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must demonstrate an absolute increase of at least 5 mm^2.
Time Frame: From randomization until documented disease progression (PD), initiation of new anti-cancer therapy, censoring date or death, whichever occurred first (up to 29 months), excluding Part 1: LGX818 300 mg group; up to 35 months for Part 1: LGX 300 mg group
Population: FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg
Number analyzed (Participants) | 192 | 194
months | 14.9 [11.0 to 18.5] | 9.6 [7.4 to 14.8]

3. Secondary Outcome: Part 2: Progression Free Survival (PFS) by BIRC in Combo 300 Group as Compared to LGX818 Group
Description: as for outcome 2
Time Frame: From randomization until documented disease progression (PD), initiation of new anti-cancer therapy, censoring date or death, whichever occurred first (up to 35 months)
Population: FAS included all randomized participants. It was planned to report combined result data of Part 1 and Part 2 for LGX818 300 mg arm.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Part 1 + Part 2: LGX818 300 mg: Participants of Part 1 and 2 received 300 mg of LGX818 orally once daily for each 28 day treatment cycle until PD as confirmed by BIRC, withdrawal of consent, intolerable toxicity, and study discontinuation, lost to follow-up or death.
Arm/Group | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 258 | 86 | 280
months | 12.9 [10.1 to 14.0] | 7.4 [5.6 to 9.2] | 9.2 [7.4 to 11.0]

4. Secondary Outcome: Part 1: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of randomization to the date of death due to any cause. If a death had not been observed by the date of analysis cutoff, OS was censored at the date of last contact.
Time Frame: From randomization until documented disease progression (PD), initiation of new anti-cancer therapy, censoring date or death, whichever occurred first (up to 38 months)
Reporting Status: Not Posted, anticipated posting 2025-08

5. Secondary Outcome: Part 1: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) as Graded by National Cancer Institute Common Terminology Criteria (NCI-CTCAE), Version 4.03
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was any untoward medical occurrence at any dose that results in death; is life-threatening; requires inpatient hospitalization/prolongation of existing hospitalization; results in persistent/significant disability/incapacity; results in congenital anomaly/birth defect or that is considered to be important medical event. As per NCI-CTCAE version 4.03, severity was graded as Grade 1: asymptomatic/mild symptoms, clinical/diagnostic observations only; Grade 2: moderate, minimal, local/noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe/medically significant but not immediately life-threatening, hospitalization/prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence; Grade 5: death. AEs of all grades were reported.
Time Frame: Baseline up to 30 days from last dose of study drug (up to 30 months), excluding Part 1: LGX818 300 mg group; up to 36 months for Part 1 LGX 300 mg group
Population: Safety analysis set included all participants who received at least one dose of study medication and have at least one valid post-baseline safety evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID
Number analyzed (Participants) | 192 | 192 | 186
percentage of participants
  Participants with AEs | 98.4 | 99.5 | 99.5
  Participants with SAEs | 34.4 | 34.9 | 37.1

6. Secondary Outcome: Part 1: Number of Participants With Clinically Notable Shift From Baseline in Laboratory Parameter Values Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE) Grade, Version 4.03
Description: Number of participants with clinically notable shift from baseline in laboratory parameter values based on national cancer institute common terminology criteria (NCI-CTCAE) grade, Version 4.03 were graded from Grades 1 to 5. Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: Moderate; minimal, local or noninvasive intervention indicated. Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death. Clinically notable shift from baseline in laboratory parameter = worsening by at least 2 grades or to >=grade 3.
Time Frame: as for outcome 5
Population: Safety analysis set included all participants who received at least one dose of study medication and have at least one valid post-baseline safety evaluation. Here, 'Number analyzed' signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID
Number analyzed (Participants) | 192 | 192 | 186
Participants
  Hemoglobin (hypo) | 19 | 11 | 13
  Prothrombin international normalized ratio increased: number analyzed (Participants) | 192 | 188 | 181
  Prothrombin international normalized ratio increased | 0 | 1 | 3
  Lymphocytes (hypo): number analyzed (Participants) | 192 | 191 | 186
  Lymphocytes (hypo) | 20 | 15 | 41
  Lymphocytes (hyper): number analyzed (Participants) | 192 | 191 | 186
  Lymphocytes (hyper) | 14 | 11 | 5
  Neutrophils (hypo) | 14 | 5 | 3
  Platelets (hypo) | 2 | 1 | 1
  Leukocytes (hypo) | 5 | 3 | 4
  Albumin (hypo) | 3 | 5 | 2
  Alkaline phosphatase | 6 | 3 | 4
  Alanine aminotransferase | 15 | 8 | 8
  Aspartate aminotransferase | 12 | 4 | 4
  Bilirubin | 1 | 0 | 13
  Creatine (phospho)kinase: number analyzed (Participants) | 186 | 182 | 180
  Creatine (phospho)kinase | 32 | 1 | 1
  Corrected Calcium (hypo): number analyzed (Participants) | 192 | 191 | 186
  Corrected Calcium (hypo) | 1 | 1 | 3
  Corrected Calcium (hyper): number analyzed (Participants) | 192 | 191 | 186
  Corrected Calcium (hyper) | 0 | 0 | 2
  Creatinine | 35 | 15 | 48
  Gamma-glutamyl transferase: number analyzed (Participants) | 192 | 191 | 186
  Gamma-glutamyl transferase | 43 | 29 | 15
  Glucose serum fasting (hypo): number analyzed (Participants) | 155 | 149 | 125
  Glucose serum fasting (hypo) | 2 | 4 | 3
  Glucose serum fasting (hyper): number analyzed (Participants) | 155 | 149 | 125
  Glucose serum fasting (hyper) | 20 | 12 | 12
  Magnesium (hypo): number analyzed (Participants) | 192 | 190 | 186
  Magnesium (hypo) | 0 | 1 | 0
  Magnesium (hyper): number analyzed (Participants) | 192 | 190 | 186
  Magnesium (hyper) | 2 | 0 | 1
  Phosphate (hypo): number analyzed (Participants) | 192 | 190 | 186
  Phosphate (hypo) | 18 | 25 | 35
  Potassium (hypo) | 1 | 1 | 3
  Potassium (hyper) | 6 | 4 | 6
  Sodium (hypo) | 7 | 1 | 1

7. Secondary Outcome: Part 1: Number of Participants With Newly Occurring Notably Abnormal Vital Signs
Description: Notably abnormal vital signs were: Low/high systolic blood pressure (SBP) (millimeter of mercury [mmHg]): less than or equal to (<=) 90 mmHg with decrease from baseline of greater than or equal to (>=) 20 mmHg/>= 160 mmHg with increase from baseline of >=20 mmHg. Low/high diastolic blood pressure (DBP) [mmHg]: <= 50 mmHg with decrease from baseline of >=15 mmHg/>=100 mmHg with increase from baseline of >=15 mmHg. Low/high Pulse rate: <=50 beats per minute (bpm) with decrease from baseline of >=15 bpm/>= 120 bpm with increase from baseline of >=15 bpm. Low/high Weight [kilogram]: >=20 percent (%) decrease from baseline/>= 10% increase from baseline. Low/high Body temperature degree Celsius (C): <= 36 degree C/>= 37.5 degree C.
Time Frame: as for outcome 5
Population: Safety analysis set included all participants who received at least one dose of study medication and have at least one valid post-baseline safety evaluation. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number analyzed" signifies participants evaluable at specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID
Number analyzed (Participants) | 188 | 185 | 184
Participants
  Sitting Pulse Rate (bpm): High: number analyzed (Participants) | 186 | 184 | 182
  Sitting Pulse Rate (bpm): High | 1 | 7 | 8
  Sitting Pulse Rate (bpm): Low: number analyzed (Participants) | 185 | 181 | 182
  Sitting Pulse Rate (bpm): Low | 3 | 8 | 2
  Sitting Systolic Blood Pressure (mmHg): High: number analyzed (Participants) | 177 | 177 | 173
  Sitting Systolic Blood Pressure (mmHg): High | 27 | 14 | 31
  Sitting Systolic Blood Pressure (mmHg): Low: number analyzed (Participants) | 188 | 184 | 182
  Sitting Systolic Blood Pressure (mmHg): Low | 7 | 4 | 1
  Sitting Diastolic Blood Pressure (mmHg): High: number analyzed (Participants) | 182 | 183 | 181
  Sitting Diastolic Blood Pressure (mmHg): High | 23 | 5 | 13
  Sitting Diastolic Blood Pressure (mmHg): Low | 9 | 7 | 5
  Weight (kg): High: number analyzed (Participants) | 187 | 184 | 184
  Weight (kg): High | 44 | 10 | 8
  Weight (kg): Low: number analyzed (Participants) | 187 | 184 | 184
  Weight (kg): Low | 2 | 8 | 13
  Body temperature (degree C): High: number analyzed (Participants) | 185 | 176 | 181
  Body temperature (degree C): High | 19 | 11 | 17
  Body temperature (degree C): Low: number analyzed (Participants) | 132 | 134 | 141
  Body temperature (degree C): Low | 76 | 74 | 57

8. Secondary Outcome: Part 1: Number of Participants With Newly Occurring Notable Electrocardiogram (ECG) Values
Description: Newly occurring notable ECG values were reported for QT (millisecond [ms]), QTcF (millisecond), QTcB (millisecond) and heart rate (beats per minute). Newly occurring was defined as participants not meeting criterion at baseline and meeting criterion post-baseline. Ranges for newly occurring notable ECG values (QT, QTcF, QTcB) are New greater than (>) 450, New >480, New >500, Increase from baseline >30, Increase from baseline >60. Heart rate: New <60, New >100 was considered as newly occurring notable value.
Time Frame: as for outcome 5
Population: Safety analysis set included all participants who received at least one dose of study medication and have at least one valid post-baseline safety evaluation. Here "Overall Number of Participants analyzed" signifies number of participants evaluable for this outcome measure and 'Number analyzed' signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID
Number analyzed (Participants) | 187 | 180 | 179
Participants
  QT: Increase >30 ms | 105 | 68 | 81
  QT: Increase >60 ms | 27 | 19 | 24
  QT: New >450 ms: number analyzed (Participants) | 180 | 169 | 173
  QT: New >450 ms | 23 | 15 | 17
  QT: New >480 ms: number analyzed (Participants) | 187 | 176 | 178
  QT: New >480 ms | 5 | 4 | 3
  QT: New >500 ms: number analyzed (Participants) | 187 | 178 | 179
  QT: New >500 ms | 2 | 2 | 2
  QTcF: Increase >30 ms: number analyzed (Participants) | 186 | 179 | 179
  QTcF: Increase >30 ms | 50 | 56 | 76
  QTcF: Increase >60 ms: number analyzed (Participants) | 186 | 179 | 179
  QTcF: Increase >60 ms | 10 | 7 | 10
  QTcF: New >450 ms: number analyzed (Participants) | 178 | 171 | 174
  QTcF: New >450 ms | 25 | 39 | 42
  QTcF: New >480 ms: number analyzed (Participants) | 186 | 177 | 179
  QTcF: New >480 ms | 7 | 7 | 5
  QTcF: New >500 ms: number analyzed (Participants) | 186 | 178 | 179
  QTcF: New >500 ms | 1 | 5 | 3
  QTcB: Increase >30 ms: number analyzed (Participants) | 184 | 179 | 177
  QTcB: Increase >30 ms | 47 | 74 | 78
  QTcB: Increase >60 ms: number analyzed (Participants) | 184 | 179 | 177
  QTcB: Increase >60 ms | 11 | 15 | 14
  QTcB: New >450 ms: number analyzed (Participants) | 155 | 158 | 155
  QTcB: New >450 ms | 47 | 76 | 65
  QTcB: New >480 ms: number analyzed (Participants) | 183 | 174 | 176
  QTcB: New >480 ms | 12 | 23 | 20
  QTcB: New >500 ms: number analyzed (Participants) | 183 | 179 | 177
  QTcB: New >500 ms | 3 | 10 | 8
  Heart rate: New <60 bpm: number analyzed (Participants) | 163 | 159 | 153
  Heart rate: New <60 bpm | 58 | 37 | 16
  Heart rate: New <100 bpm: number analyzed (Participants) | 182 | 175 | 170
  Heart rate: New <100 bpm | 14 | 23 | 18

9. Secondary Outcome: Part 1: Number of Participants With Worst Post-baseline Left Ventricular Dysfunction Events (LVEF) Values by Multigated Acquisition (MUGA) Scans or Transthoracic Echocardiograms (ECHO), by CTCAE Grade
Description: Participants with worst post-baseline LVEF Values were graded as Grade 0: Non missing value below Grade 2; Grade 2: LVEF between 40% and 50% or absolute reduction from baseline >=10% and < 20%; Grade 3: LVEF between 20% and 39% or absolute reduction from baseline >=20%; Grade 4: LVEF lower than 20%. Baseline was defined as the last non-missing value prior to the first dose of study treatment. Missing data were due to participants who died or withdrew consent prior to the first scheduled evaluation or missed evaluations as protocol deviations.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID
Number analyzed (Participants) | 192 | 192 | 186
Participants
  Grade 0 | 127 | 161 | 161
  Grade 2 | 56 | 17 | 16
  Grade 3 | 3 | 4 | 2
  Grade 4 | 0 | 0 | 0
  Missing | 6 | 10 | 7

10. Secondary Outcome: Part 1: Number of Participants With Dermatologic-related Adverse Events of Special Interest (AESI) Graded According to the National Cancer Institute Common Terminology Criteria (NCI-CTCAE) v4.03
Description: AESI consisted of events for which there was a specific clinical interest with regard to LGX818 and/or MEK162 treatment. Dermatologic-related AESI included rash, photosensitivity, nail disorders, skin infections, severe cutaneous adverse reactions and Palmar-plantar erythrodysaesthesia (PPE) syndrome. As per NCI-CTCAE version 4.03, severity was graded as Grade 1: asymptomatic/mild symptoms, clinical/diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local/noninvasive intervention indicated, limiting age-appropriate instrumental ADL; Grade 3: severe/medically significant but not immediately life-threatening, hospitalization/prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. AEs of grade 3 or 4 are reported in this outcome measure.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID
Number analyzed (Participants) | 192 | 192 | 186
Participants
  Rash | 2 | 10 | 25
  Skin infections | 4 | 1 | 0
  PPE syndrome | 0 | 26 | 2
  Photosensitivity | 1 | 0 | 3
  Nail disorders | 0 | 0 | 0
  Severe cutaneous adverse reactions | 0 | 1 | 5

11. Secondary Outcome: Part 1: Number of Participants With Ocular-related Adverse Events of Special Interest (AESI) Graded According to the National Cancer Institute Common Terminology Criteria (NCI-CTCAE) v4.03
Description: AESI consisted of events for which there was a specific clinical interest with regard to LGX818 and/or MEK162 treatment. Ocular-related AESI included retinopathy excluding retinal vein occlusion (RVO), RVO and uveitis-type events. As per NCI-CTCAE version 4.03, severity was graded as Grade 1: asymptomatic/mild symptoms, clinical/diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local/noninvasive intervention indicated, limiting age-appropriate instrumental ADL; Grade 3: severe/medically significant but not immediately life-threatening, hospitalization/prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. AEs of grade 3 or 4 are reported in this outcome measure.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID
Number analyzed (Participants) | 192 | 192 | 186
Participants
  Retinopathy excluding RVO | 5 | 0 | 0
  RVO | 0 | 1 | 0
  Uveitis-type events | 1 | 0 | 0

12. Secondary Outcome: Part 2: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) as Graded by National Cancer Institute Common Terminology Criteria (NCI-CTCAE), Version 4.03
Description: as for outcome 5
Time Frame: Baseline up to 30 days after last dose of study drug (up to 36 months)
Population: Safety analysis set included all participants who received at least one dose of study medication and have at least one valid post-baseline safety evaluation. It was planned to report combined result data of Part 1 and Part 2 for LGX818 300 mg arm.
Measure: Number; unit: percentage of Participants
Arm/Group | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 257 | 84 | 276
percentage of Participants
  AEs | 98.1 | 96.4 | 98.6
  SAEs | 29.2 | 29.8 | 33.3

13. Secondary Outcome: Part 2: Number of Participants With Clinically Notable Shift From Baseline in Laboratory Parameter Values Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE) Grade, Version 4.0
Description: Number of participants with clinically notable shift from baseline in laboratory parameter values based on national cancer institute common terminology criteria (NCI-CTCAE) grade, Version 4.0 were graded from Grades 1 to 5. Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: Moderate; minimal, local or noninvasive intervention indicated. Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death. Clinically notable shift from baseline in laboratory parameter = worsening by at least 2 grades or to >=grade 3.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 36 months)
Population: Safety analysis set included all participants who received at least one dose of study medication and have at least one valid post-baseline safety evaluation. Here, 'Number analyzed' signifies number of participants evaluable for specified rows. It was planned to report combined result data of Part 1 and Part 2 for LGX818 300 mg arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 257 | 84 | 276
Participants
  Hemoglobin (hypo) | 16 | 5 | 16
  Prothrombin international normalized ratio increased: number analyzed (Participants) | 246 | 80 | 268
  Prothrombin international normalized ratio increased | 4 | 0 | 1
  Lymphocytes (hypo): number analyzed (Participants) | 257 | 84 | 275
  Lymphocytes (hypo) | 28 | 10 | 25
  Lymphocytes (hyper): number analyzed (Participants) | 257 | 84 | 275
  Lymphocytes (hyper) | 11 | 2 | 13
  Neutrophils (hypo) | 19 | 4 | 9
  Platelets (hypo): number analyzed (Participants) | 256 | 84 | 276
  Platelets (hypo) | 1 | 1 | 2
  Leukocytes (hypo) | 3 | 2 | 5
  Albumin (hypo) | 7 | 4 | 9
  Alkaline phosphatase (hyper) | 11 | 1 | 4
  Alanine aminotransferase | 18 | 1 | 9
  Aspartate aminotransferase | 15 | 1 | 5
  Bilirubin | 2 | 0 | 0
  Creatine kinase: number analyzed (Participants) | 257 | 76 | 258
  Creatine kinase | 40 | 0 | 1
  Corrected Calcium (hypo): number analyzed (Participants) | 257 | 84 | 275
  Corrected Calcium (hypo) | 4 | 1 | 2
  Creatinine | 44 | 11 | 26
  Gamma-glutamyl transferase: number analyzed (Participants) | 257 | 84 | 275
  Gamma-glutamyl transferase | 38 | 9 | 38
  Glucose serum fasting (hypo): number analyzed (Participants) | 257 | 67 | 216
  Glucose serum fasting (hypo) | 3 | 0 | 4
  Glucose serum fasting (hyper): number analyzed (Participants) | 257 | 67 | 216
  Glucose serum fasting (hyper) | 27 | 5 | 17
  Magnesium (hypo): number analyzed (Participants) | 257 | 84 | 274
  Magnesium (hypo) | 0 | 0 | 1
  Magnesium (hyper): number analyzed (Participants) | 257 | 84 | 274
  Magnesium (hyper) | 3 | 0 | 0
  Phosphate (hypo): number analyzed (Participants) | 257 | 84 | 274
  Phosphate (hypo) | 26 | 8 | 33
  Potassium (hypo) | 2 | 0 | 1
  Potassium (hyper) | 8 | 3 | 7
  Sodium (hypo) | 4 | 2 | 3
  Sodium (hyper) | 2 | 0 | 0

14. Secondary Outcome: Part 2: Number of Participants With Newly Occurring Notably Abnormal Vital Signs
Description: Notably abnormal vital signs were: Low/high systolic blood pressure (SBP) in millimeter of mercury (mmHg): less than or equal to (<=) 90 mmHg with decrease from baseline of greater than or equal to (>=) 20 mmHg/>= 160 mmHg with increase from baseline of >=20 mmHg, Low/high diastolic blood pressure (DBP) [mmHg]: <=50 mmHg with decrease from baseline of >=15 mmHg/>=100 mmHg with increase from baseline of >=15 mmHg, Low/high pulse rate [bpm]: <=50 bpm with decrease from baseline of >=15 bpm/>=120 bpm with increase from baseline of >=15 bpm, Low/high weight (kg): >=20 % decrease from baseline/>= 10% increase from baseline Low/high Body temperature degree C): <= 36°C/>= 37.5 degree C.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 36 months)
Population: Safety analysis set included all participants who received at least one dose of study medication and have at least one valid post-baseline safety evaluation. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number analyzed" signifies participants evaluable at specified rows. It was planned to report combined result data of Part 1 and Part 2 for LGX818 300 mg arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 256 | 80 | 265
Participants
  Sitting Pulse Rate (bpm): High: number analyzed (Participants) | 252 | 78 | 262
  Sitting Pulse Rate (bpm): High | 7 | 3 | 10
  Sitting Pulse Rate (bpm): Low: number analyzed (Participants) | 254 | 77 | 258
  Sitting Pulse Rate (bpm): Low | 11 | 1 | 9
  Sitting Systolic Blood Pressure (mmHg): High: number analyzed (Participants) | 243 | 76 | 253
  Sitting Systolic Blood Pressure (mmHg): High | 40 | 3 | 17
  Sitting Systolic Blood Pressure (mmHg): Low: number analyzed (Participants) | 255 | 78 | 262
  Sitting Systolic Blood Pressure (mmHg): Low | 10 | 4 | 8
  Sitting Diastolic Blood Pressure (mmHg): High: number analyzed (Participants) | 253 | 78 | 261
  Sitting Diastolic Blood Pressure (mmHg): High | 41 | 2 | 7
  Sitting Diastolic Blood Pressure (mmHg): Low: number analyzed (Participants) | 255 | 77 | 262
  Sitting Diastolic Blood Pressure (mmHg): Low | 7 | 2 | 9
  Weight (kg): High: number analyzed (Participants) | 256 | 80 | 264
  Weight (kg): High | 46 | 1 | 11
  Weight (kg): Low: number analyzed (Participants) | 256 | 80 | 264
  Weight (kg): Low | 0 | 1 | 9
  Body temperature (°C): High: number analyzed (Participants) | 252 | 77 | 253
  Body temperature (°C): High | 14 | 5 | 16
  Body temperature (°C): Low: number analyzed (Participants) | 201 | 55 | 189
  Body temperature (°C): Low | 120 | 22 | 96

15. Secondary Outcome: Part 2: Number of Participants With Newly Occurring Notable ECG Values
Description: Newly occurring notable ECG values were reported for QT (ms), QTcF (ms), QTcB (ms) and heart rate (bpm). Newly occurring was defined as participants not meeting criterion at baseline and meeting criterion post-baseline. Ranges for newly occurring notable ECG values (QT, QTcF, QTcB) are New >450, New >480, New >500, increase from baseline >30, Increase from baseline >60. Heart rate: New < 60, New >100 was considered as newly occurring notable value.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 36 months)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 251 | 79 | 259
Participants
  QT (ms): Increase from baseline > 30 | 132 | 27 | 95
  QT (ms): Increase from baseline > 60 | 34 | 6 | 25
  QT (ms): New > 450: number analyzed (Participants) | 239 | 76 | 245
  QT (ms): New > 450 | 34 | 5 | 20
  QT (ms): New > 480: number analyzed (Participants) | 249 | 79 | 255
  QT (ms): New > 480 | 9 | 2 | 6
  QT (ms): New > 500: number analyzed (Participants) | 251 | 79 | 257
  QT (ms): New > 500 | 4 | 0 | 2
  QTcF (ms): Increase from baseline > 30: number analyzed (Participants) | 250 | 78 | 257
  QTcF (ms): Increase from baseline > 30 | 59 | 20 | 76
  QTcF (ms): Increase from baseline > 60: number analyzed (Participants) | 250 | 78 | 257
  QTcF (ms): Increase from baseline > 60 | 13 | 7 | 14
  QTcF (ms): New > 450: number analyzed (Participants) | 240 | 70 | 241
  QTcF (ms): New > 450 | 36 | 11 | 50
  QTcF (ms): New > 480: number analyzed (Participants) | 249 | 78 | 255
  QTcF (ms): New > 480 | 11 | 5 | 12
  QTcF (ms): New > 500: number analyzed (Participants) | 250 | 78 | 256
  QTcF (ms): New > 500 | 2 | 1 | 6
  QTcB (ms): New > 450: number analyzed (Participants) | 216 | 67 | 225
  QTcB (ms): New > 450 | 70 | 28 | 104
  QTcB (ms): New > 480: number analyzed (Participants) | 247 | 77 | 251
  QTcB (ms): New > 480 | 23 | 6 | 29
  QTcB (ms): New > 500: number analyzed (Participants) | 250 | 79 | 258
  QTcB (ms): New > 500 | 10 | 1 | 11
  QTcB (ms): Increase from baseline > 30: number analyzed (Participants) | 250 | 79 | 258
  QTcB (ms): Increase from baseline > 30 | 69 | 24 | 98
  QTcB (ms): Increase from baseline > 60: number analyzed (Participants) | 250 | 79 | 258
  QTcB (ms): Increase from baseline > 60 | 22 | 8 | 23
  Heart rate (bpm): New < 60: number analyzed (Participants) | 213 | 67 | 226
  Heart rate (bpm): New < 60 | 82 | 5 | 42
  Heart rate (bpm): New > 100: number analyzed (Participants) | 241 | 74 | 249
  Heart rate (bpm): New > 100 | 8 | 10 | 33

16. Secondary Outcome: Part 2: Number of Participants With Worst Post-baseline Left Ventricular Dysfunction Events (LVEF) Values by Multigated Acquisition (MUGA) Scans or Transthoracic Echocardiograms (ECHO), by CTCAE Grade
Description: Participants with worst post-baseline LVEF Values were graded as Grade 0: Non missing value below Grade 2; Grade 2: LVEF between 40% and 50% or absolute reduction from baseline >=10% and < 20%;Grade 3: LVEF between 20% and 39% or absolute reduction from baseline >=20%; Grade 4: LVEF lower than 20%. Baseline was defined as the last non-missing value prior to the first dose of study treatment. Missing data were due to participants who died or withdrew consent prior to the first scheduled evaluation or missed evaluations as protocol deviations.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 36 months)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 257 | 84 | 276
Participants
  Grade 0 | 181 | 74 | 235
  Grade 2 | 71 | 5 | 22
  Grade 3 | 3 | 0 | 4
  Grade 4 | 0 | 0 | 0
  Missing | 2 | 5 | 15

17. Secondary Outcome: Part 2: Number of Participants With Dermatologic-related Adverse Events of Special Interest (AESI) Graded According to the National Cancer Institute Common Terminology Criteria (NCI-CTCAE) v4.03
Description: AESI consisted of events for which there was a specific clinical interest with regard to LGX818 and/or MEK162 treatment. Dermatologic-related AESI included rash, photosensitivity, nail disorders, skin infections, severe cutaneous adverse reactions and PPE syndrome. As per NCI-CTCAE version 4.03, severity was graded as Grade 1: asymptomatic/mild symptoms, clinical/diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local/noninvasive intervention indicated, limiting age-appropriate instrumental ADL; Grade 3: severe/medically significant but not immediately life-threatening, hospitalization/prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. AEs of grade 3 or 4 are reported are reported in this outcome measure.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 36 months)
Population: Safety analysis set includes all participants who received at least one dose of study medication and have at least one valid post-baseline safety evaluation. It was planned to report combined result data of Part 1 and Part 2 for LGX818 300 mg arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 257 | 84 | 276
Participants
  Rash | 2 | 3 | 13
  Skin infection | 7 | 0 | 1
  PPE syndrome | 1 | 4 | 30
  Photosensitivity | 0 | 0 | 0
  Nail disorders | 0 | 0 | 0
  Severe cutaneous adverse reactions | 0 | 0 | 1

18. Secondary Outcome: Part 2: Number of Participants With Ocular-related Adverse Events of Special Interest (AESI) Graded According to the National Cancer Institute Common Terminology Criteria (NCI-CTCAE) v4.03
Description: AESI consisted of events for which there was a specific clinical interest with regard to LGX818 and/or MEK162 treatment. Ocular-related AESI included retinopathy excluding RVO, RVO and uveitis-type events. As per NCI-CTCAE version 4.03, severity was graded as Grade 1: asymptomatic/mild symptoms, clinical/diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local/noninvasive intervention indicated, limiting age-appropriate instrumental ADL; Grade 3: severe/medically significant but not immediately life-threatening, hospitalization/prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. AEs of grade 3 or 4 are reported in this outcome measure.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 36 months)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 257 | 84 | 276
Participants
  Retinopathy excluding RVO | 4 | 0 | 0
  RVO | 0 | 0 | 1
  Uveitis-type events | 4 | 0 | 0

19. Secondary Outcome: Part 2: Overall Survival (OS)
Time Frame: as for outcome 4
Reporting Status: Not Posted, anticipated posting 2025-08

20. Secondary Outcome: Part 1 and Part 2: Objective Response Rate (ORR)
Description: ORR, calculated as the percentage of participants with a best overall response of complete response (CR) or partial response (PR). CR was defined as disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. Results are reported for confirmed BIRC response.
Time Frame: From randomization until disease progression, censoring date or death, whichever occurred first (up to 29 months for Part 1, excluding Part 1: LGX818 300 mg group; up to 35 months for Part 2 and Part 1 LGX 300 mg group)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 192 | 194 | 191 | 258 | 86 | 280
percentage of participants | 63.0 [55.8 to 69.9] | 50.5 [43.3 to 57.8] | 40.3 [33.3 to 47.6] | 65.9 [59.8 to 71.7] | 50.0 [39.0 to 61.0] | 50.4 [44.3 to 56.4]

21. Secondary Outcome: Part 1 and Part 2: Time to Objective Response (TTR)
Description: TTR was the time between date of randomization until first documented response of CR or PR. Participants who did not achieve a PR or CR were censored at the last adequate tumor assessment date when they did not have a PFS event or at maximum follow-up (i.e. first patient first visit [FPFV] to last patient last visit [LPLV] used for the analysis) when they had a PFS event. CR was defined as disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. TTR was estimated in the treatment arms using a Kaplan-Meier method. TTR was based on central review.
Time Frame: as for outcome 20
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 192 | 194 | 191 | 258 | 86 | 280
months | 1.9 [1.9 to 1.9] | 2.0 [1.9 to 3.6] | 2.1 [1.9 to 3.7] | 1.9 [1.9 to 2.0] | 1.9 [1.9 to 2.3] | 1.9 [1.9 to 3.2]

22. Secondary Outcome: Part 1 and Part 2: Disease Control Rate (DCR)
Description: DCR was calculated as the percentage of participants with a best overall response (BOR) of CR, PR, or stable disease (SD). CR was defined as disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. Two sets of DCR were considered, one for confirmed and one for unconfirmed responses. Results are reported for confirmed and unconfirmed responses combined. SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD. DCR was based on central review.
Time Frame: From randomization until disease progression or death, whichever occurred first (up to 29 months for Part 1, excluding Part 1: LGX818 300 mg group; up to 35 months for Part 2 and Part 1 LGX 300 mg group)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 192 | 194 | 191 | 258 | 86 | 280
percentage of participants | 92.2 [87.4 to 95.6] | 84.0 [78.1 to 88.9] | 81.7 [75.4 to 86.9] | 90.7 [86.5 to 93.9] | 79.1 [69.0 to 87.1] | 82.5 [77.5 to 86.8]

23. Secondary Outcome: Part 1 and Part 2: Duration of Response (DOR)
Description: DOR was calculated, as the time from the date of first documented response (CR or PR) to the first documented progression or death due to underlying cancer. DOR was estimated for responders (i.e. participants achieving at least once CR or PR) only using a Kaplan-Meier method. CR was defined as disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. If a participant with a CR or PR had no progression or death due to underlying disease, the participant was censored at the date of last adequate tumor assessment. Results are based on confirmed BIRC response.
Time Frame: as for outcome 20
Population: Analysis population included all the participants who achieved at least once confirmed CR or PR. It was planned to report combined result data of Part 1 and Part 2 for LGX818 300 mg arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 121 | 98 | 77 | 170 | 43 | 141
months | 16.6 [12.2 to 20.4] | 15.2 [11.1 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | 12.3 [6.9 to 16.9] | 12.7 [9.3 to 15.1] | 7.5 [5.6 to 14.0] | 12.9 [8.9 to 15.5]

24. Secondary Outcome: Part 1 and Part 2: Time to Definitive 10% Deterioration in the Function Assessment Cancer Therapy-melanoma (FACT-M) Subscale
Description: FACT-M:melanoma specific questionnaire to assess participant health-related quality of life. Melanoma specific subscale consists of 16 items related to signs,symptoms,physical/social activities most relevant to participants with advanced-stage melanoma. Other items include physical, functional and social/family well-being (7 items each),emotional well-being (6 items),surgery specific concerns related to melanoma(8 items,not included in this study). Each item range from 0(not at all) to 4(very much), combined to produce subscale scores.Total score range for FACT-M excluding surgery specific items is 0 to 172,higher scores represent better quality of life.Melanoma subscale score range from 0(worst response) to 64(best response),higher score indicated better quality of life. Time to definitive 10% deterioration:time from date of randomization to date of event with at least 10% relative to baseline worsening of corresponding scale score with no later improvement or death due to any cause.
Time Frame: Date of randomization to date of event or death due to any cause, which ever occurred first (up to 29 months for Part 1, excluding Part 1: LGX818 300 mg group; up to 35 months for Part 2 and Part 1 LGX 300 mg group)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 192 | 194 | 191 | 258 | 86 | 280
months | NA [22.1 to NA] — Median and upper limit of 95% CI were not estimable due to low number of participants with events. | 30.5 [18.4 to 30.5] | 22.1 [15.2 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | NA [NA to NA] — Median and 95% CI were not estimable due to low number of participants with events. | NA [9.4 to NA] — Median and upper limit of 95% CI were not estimable due to low number of participants with events. | 20.5 [16.6 to 30.5]

25. Secondary Outcome: Part 1 and Part 2: Time to Definitive 10% Deterioration in the Global Health Status Score of the European Organization for Research and Treatment of Cancer's Core Quality of Life Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is 30 item questionnaire composed of 5 multi-item functional subscales (physical, role, cognitive, emotional, social functioning), 3 multi-item symptom scales (fatigue, nausea/vomiting, and pain), global health/quality of life (QOL) subscale and 6 single items assessing other cancer related symptoms (dyspnea, sleep disturbance, appetite, diarrhea, constipation and financial impact of cancer). It employed twenty-eight 4 point Likert scales with responses from "not at all" to "very much" and two 7 point Likert scales for global health and overall QOL. Global health status scale score ranged from 0 to 100. Higher score represented better level of functioning. Time to definitive 10% deterioration: time from date of randomization to date of event with at least 10% relative to baseline worsening of corresponding scale score with no later improvement or death due to any cause.
Time Frame: Date of randomization to date of event or death due to any cause, which ever occurred first (maximum up to 29 months for Part 1, excluding Part 1: LGX818 300 mg group; up to 35 months for Part 2 and Part 1 LGX 300 mg group)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 192 | 194 | 191 | 258 | 86 | 280
months | 23.9 [20.4 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | 14.7 [8.1 to 24.0] | 16.6 [11.9 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | 18.4 [16.8 to 19.1] | 9.5 [5.6 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | 11.1 [7.7 to 20.2]

26. Secondary Outcome: Part 1 and Part 2: Change From Baseline in the Function Assessment Cancer Therapy-melanoma (FACT-M) Subscale at Day 1 of Cycle 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25 and End of Treatment Visit
Description: FACT-M: melanoma specific questionnaire to assess participant health-related quality of life. Melanoma specific subscale consists of 16 items related to signs, symptoms, physical/social activities most relevant to participants with advanced-stage melanoma. Other items include physical, functional and social/family well-being (7 items each),emotional well-being (6 items),surgery specific concerns related to melanoma(8 items, not included in this study). Each item range from 0(not at all) to 4(very much), combined to produce subscale scores. Total score range for FACT-M excluding surgery specific items is 0 to 172,higher scores represented better quality of life. Melanoma subscale score range from 0(worst response) to 64(best response),higher score indicated better quality of life.
Time Frame: Baseline (Day 1 of Cycle 1), Day 1 of Cycle 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25 and end of treatment visit (within14 days after the last dose of study drug)
Population: FAS included all randomized participants. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number analyzed" signifies participants evaluable for each specified row. It was planned to report combined result data of Part 1 and Part 2 for LGX818 300 mg arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 165 | 177 | 159 | 234 | 83 | 260
units on a scale
  Baseline | 52.39 (9.053) | 52.76 (8.206) | 52.01 (8.650) | 52.08 (8.493) | 51.13 (9.567) | 52.24 (8.679)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 141 | 148 | 128 | 212 | 67 | 215
  Change at Cycle 3 Day 1 | 0.92 (9.539) | -3.58 (8.133) | -1.55 (9.023) | 2.79 (7.296) | -2.16 (9.700) | -3.14 (8.654)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 128 | 132 | 106 | 200 | 60 | 192
  Change at Cycle 5 Day 1 | -0.01 (9.157) | -3.77 (7.576) | -1.90 (7.572) | 2.58 (7.244) | -0.60 (7.948) | -2.78 (7.814)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 120 | 109 | 84 | 177 | 52 | 161
  Change at Cycle 7 Day 1 | 1.35 (9.595) | -3.05 (6.633) | -2.19 (8.651) | 2.64 (7.766) | -3.14 (9.559) | -3.08 (7.670)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 103 | 79 | 63 | 161 | 41 | 120
  Change at Cycle 9 Day 1 | 0.52 (9.096) | -2.69 (6.513) | -1.90 (7.491) | 3.23 (7.720) | -1.83 (7.323) | -2.39 (6.782)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 87 | 72 | 46 | 143 | 31 | 103
  Change at Cycle 11 Day 1 | 0.18 (7.768) | -3.67 (6.418) | -0.51 (7.436) | 2.54 (7.796) | -2.41 (7.653) | -3.29 (6.800)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 77 | 65 | 39 | 126 | 26 | 91
  Change at Cycle 13 Day 1 | -0.33 (8.855) | -2.71 (7.187) | -0.97 (8.818) | 1.97 (8.127) | -3.31 (7.902) | -2.88 (7.359)
  Change at Cycle 15 Day 1: number analyzed (Participants) | 68 | 56 | 29 | 95 | 18 | 74
  Change at Cycle 15 Day 1 | 0.40 (7.943) | -2.48 (6.829) | -1.72 (9.906) | 2.08 (9.196) | -4.14 (5.662) | -2.88 (6.566)
  Change at Cycle 17 Day 1: number analyzed (Participants) | 58 | 50 | 23 | 64 | 14 | 64
  Change at Cycle 17 Day 1 | 0.27 (7.775) | -1.66 (6.681) | 0.70 (6.071) | 2.45 (9.012) | -2.64 (9.724) | -1.88 (7.375)
  Change at Cycle 19 Day 1: number analyzed (Participants) | 47 | 51 | 20 | 26 | 9 | 60
  Change at Cycle 19 Day 1 | -0.59 (7.257) | -2.80 (6.172) | 0.23 (9.094) | 1.23 (10.618) | 0.00 (11.467) | -2.38 (7.150)
  Change at Cycle 21 Day 1: number analyzed (Participants) | 33 | 39 | 15 | 12 | 1 | 40
  Change at Cycle 21 Day 1 | -0.69 (6.947) | -2.59 (6.528) | -3.33 (6.399) | 2.58 (8.218) | -2.00 | -2.58 (6.445)
  Change at Cycle 23 Day 1: number analyzed (Participants) | 22 | 34 | 12 | 0 | 0 | 34
  Change at Cycle 23 Day 1 | -1.67 (7.003) | -1.38 (6.818) | -0.17 (4.687) |  |  | -1.38 (6.818)
  Change at Cycle 25 Day 1: number analyzed (Participants) | 18 | 25 | 7 | 0 | 0 | 25
  Change at Cycle 25 Day 1 | -1.83 (6.205) | -1.00 (6.880) | -0.14 (5.305) |  |  | -1.00 (6.880)
  Change at End of treatment visit: number analyzed (Participants) | 2 | 8 | 7 | 6 | 5 | 13
  Change at End of treatment visit | 18.50 (23.335) | -5.18 (11.458) | -2.31 (4.715) | 6.58 (7.197) | -1.61 (9.115) | -3.81 (10.370)

27. Secondary Outcome: Part 1 and Part 2: Change From Baseline in EuroQoL-5 Dimension-5 Level (EQ-5D-5L) Index Score at Day 1 of Cycle 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25 and End of Treatment Visit
Description: EQ-5D-5L is a standardized participant completed questionnaire that measures health status in terms of a single index value or utility score. EQ-5D-5L consisted of two components: a health state profile (descriptive system) and a visual analogue scale (VAS) in which participants rate their overall health status from 0 (worst imaginable) to 100 (best imaginable), where higher scores indicated better health status. EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 response levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. EQ-5D-5L health status index score range between 0 to 1. Higher score indicated better health status.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 167 | 181 | 161 | 235 | 83 | 264
units on a scale
  Baseline | 0.74 (0.210) | 0.76 (0.181) | 0.73 (0.222) | 0.75 (0.219) | 0.73 (0.244) | 0.75 (0.203)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 153 | 157 | 143 | 224 | 67 | 224
  Change at Cycle 3 Day 1 | 0.05 (0.194) | -0.10 (0.199) | 0.00 (0.196) | 0.06 (0.204) | -0.06 (0.246) | -0.09 (0.214)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 136 | 139 | 116 | 206 | 59 | 198
  Change at Cycle 5 Day 1 | 0.04 (0.196) | -0.15 (0.220) | -0.04 (0.196) | 0.07 (0.218) | -0.06 (0.231) | -0.13 (0.227)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 125 | 116 | 88 | 187 | 53 | 169
  Change at Cycle 7 Day 1 | 0.05 (0.201) | -0.13 (0.189) | -0.03 (0.215) | 0.06 (0.237) | -0.16 (0.220) | -0.14 (0.199)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 114 | 87 | 68 | 163 | 43 | 130
  Change at Cycle 9 Day 1 | 0.03 (0.237) | -0.15 (0.197) | -0.04 (0.237) | 0.07 (0.192) | -0.11 (0.202) | -0.14 (0.199)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 95 | 72 | 50 | 144 | 33 | 105
  Change at Cycle 11 Day 1 | 0.04 (0.197) | -0.18 (0.206) | -0.01 (0.238) | 0.06 (0.195) | -0.16 (0.230) | -0.17 (0.213)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 79 | 63 | 40 | 130 | 27 | 90
  Change at Cycle 13 Day 1 | 0.05 (0.225) | -0.17 (0.206) | -0.02 (0.263) | 0.05 (0.254) | -0.20 (0.216) | -0.18 (0.208)
  Change at Cycle 15 Day 1: number analyzed (Participants) | 69 | 61 | 29 | 101 | 17 | 78
  Change at Cycle 15 Day 1 | 0.05 (0.208) | -0.18 (0.203) | -0.07 (0.280) | 0.05 (0.259) | -0.26 (0.262) | -0.20 (0.218)
  Change at Cycle 17 Day 1: number analyzed (Participants) | 60 | 56 | 25 | 66 | 12 | 68
  Change at Cycle 17 Day 1 | 0.07 (0.193) | -0.14 (0.165) | -0.02 (0.173) | 0.06 (0.188) | -0.20 (0.332) | -0.15 (0.203)
  Change at Cycle 19 Day 1: number analyzed (Participants) | 49 | 51 | 22 | 28 | 9 | 60
  Change at Cycle 19 Day 1 | 0.03 (0.239) | -0.18 (0.235) | -0.02 (0.214) | 0.05 (0.231) | -0.11 (0.328) | -0.17 (0.249)
  Change at Cycle 21 Day 1: number analyzed (Participants) | 35 | 42 | 16 | 12 | 1 | 43
  Change at Cycle 21 Day 1 | 0.07 (0.132) | -0.14 (0.198) | -0.04 (0.159) | 0.12 (0.174) | -0.11 | -0.14 (0.196)
  Change at Cycle 23 Day 1: number analyzed (Participants) | 24 | 33 | 11 | 0 | 0 | 33
  Change at Cycle 23 Day 1 | 0.04 (0.139) | -0.11 (0.147) | -0.05 (0.171) |  |  | -0.11 (0.147)
  Change at Cycle 25 Day 1: number analyzed (Participants) | 16 | 26 | 5 | 0 | 0 | 26
  Change at Cycle 25 Day 1 | 0.07 (0.135) | -0.11 (0.207) | -0.17 (0.221) |  |  | -0.11 (0.207)
  Change at End of treatment visit: number analyzed (Participants) | 3 | 5 | 3 | 5 | 4 | 9
  Change at End of treatment visit | 0.03 (0.081) | -0.09 (0.347) | -0.14 (0.103) | -0.27 (0.481) | -0.06 (0.061) | -0.08 (0.249)

28. Secondary Outcome: Part 1 and Part 2: Change From Baseline in Global Health Status Score of EORTC QLQ-C30 at Day 1 of Cycle 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25 and End of Treatment Visit
Description: EORTC QLQ-C30 contains 30 items and is composed of multi-item and single-item measures. These include 5 functional scales (physical, role, emotional, cognitive and social functioning), 3 symptom scales (fatigue, nausea/vomiting, and pain), 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial impact) and a global health status/quality of life (QOL) scale. The questionnaire employs 28 4-point Likert scales with responses from "not at all" to "very much" and two 7-point Likert scales for global health and overall QOL. Responses to all items converted to 0 to 100 scale. For functional and global QOL scales, higher scores represent a better level of functioning/QOL. For symptom-oriented scales, a higher score represents more severe symptoms.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 166 | 181 | 160 | 231 | 81 | 262
units on a scale
  Baseline | 66.72 (21.585) | 66.07 (21.890) | 64.74 (23.611) | 65.95 (23.028) | 67.39 (22.095) | 66.48 (21.920)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 152 | 156 | 135 | 220 | 69 | 225
  Change at Cycle 3 Day 1 | 3.56 (22.463) | -7.64 (21.564) | -3.46 (25.235) | 4.47 (23.031) | -4.95 (20.378) | -6.81 (21.199)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 134 | 138 | 111 | 205 | 60 | 198
  Change at Cycle 5 Day 1 | 1.55 (23.441) | -9.24 (21.611) | -4.05 (23.700) | 5.61 (19.396) | -4.72 (22.776) | -7.87 (22.011)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 125 | 114 | 85 | 188 | 53 | 167
  Change at Cycle 7 Day 1 | 1.53 (23.220) | -9.21 (23.528) | -3.04 (28.197) | 5.01 (24.000) | -7.08 (20.955) | -8.53 (22.701)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 107 | 88 | 66 | 157 | 42 | 130
  Change at Cycle 9 Day 1 | -0.55 (25.500) | -12.03 (19.771) | -6.94 (21.512) | 4.94 (20.258) | -8.73 (18.945) | -10.96 (19.496)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 71 | 46 | 147 | 31 | 102
  Change at Cycle 11 Day 1 | 0.81 (21.670) | -11.27 (20.611) | -3.80 (22.202) | 4.76 (21.212) | -7.53 (19.288) | -10.13 (20.197)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 79 | 64 | 37 | 126 | 26 | 90
  Change at Cycle 13 Day 1 | 0.42 (22.642) | -8.59 (22.516) | -2.93 (20.621) | 5.89 (23.642) | -9.29 (24.645) | -8.80 (23.013)
  Change at Cycle 15 Day 1: number analyzed (Participants) | 68 | 58 | 29 | 101 | 17 | 75
  Change at Cycle 15 Day 1 | 5.02 (19.108) | -9.91 (23.490) | -10.34 (29.852) | 6.11 (21.695) | -12.75 (21.270) | -10.56 (22.897)
  Change at Cycle 17 Day 1: number analyzed (Participants) | 61 | 55 | 24 | 64 | 14 | 69
  Change at Cycle 17 Day 1 | 0.41 (21.807) | -8.03 (17.784) | -6.94 (20.214) | 5.86 (21.806) | -7.14 (20.111) | -7.85 (18.127)
  Change at Cycle 19 Day 1: number analyzed (Participants) | 49 | 50 | 22 | 27 | 9 | 59
  Change at Cycle 19 Day 1 | -0.51 (17.547) | -9.33 (19.169) | -1.89 (20.401) | 1.23 (18.155) | -0.93 (12.805) | -8.05 (18.503)
  Change at Cycle 21 Day 1: number analyzed (Participants) | 34 | 43 | 16 | 11 | 1 | 44
  Change at Cycle 21 Day 1 | 0.74 (16.838) | -11.05 (21.725) | -8.85 (11.968) | 3.03 (19.816) | 0.00 | -10.80 (21.535)
  Change at Cycle 23 Day 1: number analyzed (Participants) | 24 | 34 | 12 | 0 | 0 | 34
  Change at Cycle 23 Day 1 | -1.39 (13.157) | -5.64 (19.754) | -3.47 (18.278) |  |  | -5.64 (19.754)
  Change at Cycle 25 Day 1: number analyzed (Participants) | 17 | 26 | 7 | 0 | 0 | 26
  Change at Cycle 25 Day 1 | 1.96 (13.349) | -7.05 (18.057) | -2.38 (19.670) |  |  | -7.05 (18.057)
  Change at End of treatment visit: number analyzed (Participants) | 2 | 7 | 4 | 4 | 2 | 9
  Change at End of treatment visit | 0.00 (11.785) | 4.76 (28.810) | -4.17 (10.758) | -6.25 (18.478) | 4.17 (29.463) | 4.63 (27.039)

29. Secondary Outcome: Part 1 and Part 2: Change From Baseline in Emotional Functioning Scale Score of the EORTC QLQ-C30 at Day 1 of Cycle 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25 and End of Treatment Visit
Description: EORTC QLQ-C30 contains 30 items and is composed of multi-item and single-item measures. These include 5 functional scales (physical, role, emotional, cognitive and social functioning), 3 symptom scales (fatigue, nausea/vomiting, and pain), 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial impact) and a global health status/quality of life (QOL) scale. The questionnaire employs 28 4-point Likert scales with responses from "not at all" to "very much" and two 7-point Likert scales for global health and overall QOL. Responses to all items converted to 0 to 100 scale. For functional and global QOL scales, higher scores represent a better level of functioning/QOL. For symptom-oriented scales, a higher score represented more severe symptoms.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 166 | 181 | 160 | 231 | 83 | 264
units on a scale
  Baseline | 74.68 (21.233) | 74.46 (22.367) | 72.31 (24.695) | 73.04 (24.450) | 74.20 (21.488) | 74.38 (22.054)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 152 | 156 | 136 | 220 | 70 | 226
  Change at Cycle 3 Day 1 | 3.23 (20.588) | -0.34 (22.138) | 1.88 (20.610) | 7.29 (20.011) | 1.79 (19.958) | 0.32 (21.465)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 134 | 139 | 111 | 205 | 62 | 201
  Change at Cycle 5 Day 1 | 5.37 (19.243) | 1.54 (22.418) | 2.03 (20.662) | 6.15 (21.401) | 2.96 (20.473) | 1.98 (21.796)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 125 | 115 | 85 | 188 | 53 | 168
  Change at Cycle 7 Day 1 | 5.42 (20.027) | 0.34 (23.104) | 2.71 (20.875) | 9.37 (21.088) | -3.62 (19.441) | -0.91 (22.033)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 107 | 88 | 67 | 157 | 42 | 130
  Change at Cycle 9 Day 1 | 4.47 (24.341) | 2.15 (19.735) | -0.17 (24.283) | 9.22 (21.940) | -0.60 (16.296) | 1.26 (18.674)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 93 | 71 | 46 | 147 | 31 | 102
  Change at Cycle 11 Day 1 | 4.81 (22.102) | 0.12 (22.205) | 4.53 (18.148) | 10.56 (20.850) | -2.69 (17.793) | -0.74 (20.915)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 79 | 64 | 37 | 126 | 26 | 90
  Change at Cycle 13 Day 1 | 3.52 (23.715) | 3.78 (19.694) | -2.25 (22.192) | 8.66 (21.894) | -6.41 (17.998) | 0.83 (19.675)
  Change at Cycle 15 Day 1: number analyzed (Participants) | 68 | 58 | 29 | 101 | 17 | 75
  Change at Cycle 15 Day 1 | 7.35 (21.813) | 2.30 (20.755) | -5.46 (26.190) | 10.59 (19.609) | -2.12 (13.232) | 1.30 (19.317)
  Change at Cycle 17 Day 1: number analyzed (Participants) | 61 | 55 | 24 | 64 | 14 | 69
  Change at Cycle 17 Day 1 | 5.33 (20.584) | 3.64 (21.502) | -1.39 (15.862) | 10.33 (20.415) | 1.79 (15.736) | 3.26 (20.373)
  Change at Cycle 19 Day 1: number analyzed (Participants) | 49 | 50 | 22 | 27 | 9 | 59
  Change at Cycle 19 Day 1 | 4.25 (19.552) | 1.00 (24.493) | 0.38 (16.158) | 8.33 (22.997) | 2.78 (16.667) | 1.27 (23.357)
  Change at Cycle 21 Day 1: number analyzed (Participants) | 34 | 43 | 16 | 11 | 1 | 44
  Change at Cycle 21 Day 1 | 4.17 (19.811) | -1.16 (23.751) | -3.13 (16.908) | 13.13 (15.619) | 16.67 | -0.76 (23.626)
  Change at Cycle 23 Day 1: number analyzed (Participants) | 24 | 34 | 12 | 0 | 0 | 34
  Change at Cycle 23 Day 1 | -1.74 (21.420) | 2.94 (22.556) | -0.69 (23.693) |  |  | 2.94 (22.556)
  Change at Cycle 25 Day 1: number analyzed (Participants) | 17 | 26 | 7 | 0 | 0 | 26
  Change at Cycle 25 Day 1 | 3.92 (11.456) | -0.32 (24.093) | -1.19 (34.503) |  |  | -0.32 (24.093)
  Change at End of treatment visit: number analyzed (Participants) | 2 | 7 | 4 | 4 | 3 | 10
  Change at End of treatment visit | 41.67 (11.785) | -3.57 (25.394) | 12.50 (28.464) | -4.17 (14.434) | 5.56 (4.811) | -0.83 (21.318)

30. Secondary Outcome: Part 1 and Part 2: Change From Baseline in Physical Functioning Scale Score of the EORTC QLQ-C30 at Day 1 of Cycle 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25 and End of Treatment Visit
Description: EORTC QLQ-C30 contains 30 items and is composed of multi-item and single-item measures. These include 5 functional scales (physical, role, emotional, cognitive and social functioning), 3 symptom scales (fatigue, nausea/vomiting, and pain), 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial impact) and a global health status/quality of life (QOL) scale. The questionnaire employs 28 4-point Likert scales with responses from "not at all" to "very much" and two 7-point Likert scales for global health and overall QOL. Responses to all items converted to 0 to 100 scale. For functional and global QOL scales, higher scores represented a better level of functioning/QOL. For symptom-oriented scales, a higher score represented more severe symptoms.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 167 | 180 | 159 | 235 | 83 | 263
units on a scale
  Baseline | 82.10 (19.593) | 83.18 (20.266) | 80.71 (22.182) | 80.67 (21.889) | 81.45 (21.890) | 82.63 (20.766)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 153 | 157 | 135 | 222 | 70 | 227
  Change at Cycle 3 Day 1 | 0.20 (18.033) | -13.79 (20.396) | -2.90 (20.319) | 2.94 (16.831) | -13.63 (22.428) | -13.74 (20.994)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 135 | 138 | 111 | 208 | 62 | 200
  Change at Cycle 5 Day 1 | 0.15 (18.388) | -17.14 (22.276) | -7.45 (17.792) | 2.73 (17.748) | -12.63 (21.570) | -15.74 (22.104)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 127 | 115 | 84 | 191 | 53 | 168
  Change at Cycle 7 Day 1 | -1.93 (18.071) | -16.26 (21.719) | -6.98 (19.605) | 1.22 (17.469) | -17.01 (20.200) | -16.49 (21.194)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 110 | 88 | 66 | 160 | 42 | 130
  Change at Cycle 9 Day 1 | -0.45 (20.511) | -19.43 (20.755) | -6.82 (21.881) | 3.03 (16.525) | -15.83 (16.269) | -18.27 (19.429)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 94 | 71 | 45 | 148 | 31 | 102
  Change at Cycle 11 Day 1 | -0.85 (18.767) | -22.65 (20.867) | -4.11 (18.680) | 0.50 (17.734) | -13.49 (13.665) | -19.87 (19.369)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 80 | 64 | 36 | 127 | 26 | 90
  Change at Cycle 13 Day 1 | -1.25 (19.705) | -20.00 (20.874) | -6.30 (22.534) | 0.47 (18.290) | -13.85 (17.781) | -18.22 (20.127)
  Change at Cycle 15 Day 1: number analyzed (Participants) | 69 | 58 | 30 | 101 | 17 | 75
  Change at Cycle 15 Day 1 | 0.29 (17.356) | -20.26 (21.030) | -6.22 (21.580) | -0.40 (22.466) | -24.31 (22.845) | -21.18 (21.364)
  Change at Cycle 17 Day 1: number analyzed (Participants) | 63 | 55 | 25 | 66 | 14 | 69
  Change at Cycle 17 Day 1 | -0.03 (17.862) | -18.88 (20.072) | -3.27 (19.817) | -0.88 (16.432) | -19.05 (23.367) | -18.91 (20.599)
  Change at Cycle 19 Day 1: number analyzed (Participants) | 49 | 49 | 21 | 28 | 9 | 58
  Change at Cycle 19 Day 1 | -1.22 (16.140) | -20.07 (21.417) | -1.90 (20.237) | -5.71 (16.301) | -14.07 (14.699) | -19.14 (20.527)
  Change at Cycle 21 Day 1: number analyzed (Participants) | 35 | 43 | 16 | 11 | 1 | 44
  Change at Cycle 21 Day 1 | -0.95 (13.150) | -16.86 (19.694) | -4.90 (19.355) | -8.48 (23.303) | -13.33 | -16.78 (19.471)
  Change at Cycle 23 Day 1: number analyzed (Participants) | 24 | 34 | 12 | 0 | 0 | 34
  Change at Cycle 23 Day 1 | -5.00 (13.656) | -14.46 (18.298) | -2.22 (19.557) |  |  | -14.46 (18.298)
  Change at Cycle 25 Day 1: number analyzed (Participants) | 17 | 25 | 7 | 0 | 0 | 25
  Change at Cycle 25 Day 1 | -5.49 (14.575) | -15.93 (17.092) | -4.76 (23.637) |  |  | -15.93 (17.092)
  Change at End of treatment visit: number analyzed (Participants) | 2 | 7 | 4 | 4 | 3 | 10
  Change at End of treatment visit | 33.33 (47.140) | -0.95 (22.910) | -15.00 (19.149) | -5.00 (10.000) | -4.44 (3.849) | -2.00 (18.869)

31. Secondary Outcome: Part 1 and Part 2: Change From Baseline in Social Functioning Scale Score of the EORTC QLQ-C30 at Day 1 of Cycle 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25 and End of Treatment Visit
Description: as for outcome 30
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 164 | 179 | 160 | 229 | 83 | 262
units on a scale
  Baseline | 80.69 (24.696) | 80.91 (23.841) | 78.54 (26.854) | 81.37 (25.262) | 78.31 (28.600) | 80.09 (25.418)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 152 | 155 | 136 | 218 | 70 | 225
  Change at Cycle 3 Day 1 | -0.66 (27.854) | -10.86 (28.967) | -4.90 (30.097) | 4.05 (22.461) | -10.00 (26.829) | -10.59 (28.262)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 133 | 137 | 111 | 203 | 62 | 199
  Change at Cycle 5 Day 1 | 3.26 (27.559) | -11.92 (32.145) | -7.21 (27.026) | 3.37 (20.604) | -5.11 (28.244) | -9.80 (31.073)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 124 | 114 | 85 | 186 | 54 | 168
  Change at Cycle 7 Day 1 | 2.82 (28.807) | -9.80 (28.979) | -2.75 (31.586) | 3.05 (22.185) | -13.89 (27.992) | -11.11 (28.646)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 106 | 87 | 67 | 155 | 42 | 129
  Change at Cycle 9 Day 1 | 1.57 (31.834) | -15.71 (26.579) | -1.99 (30.084) | 3.66 (21.002) | -9.52 (14.790) | -13.70 (23.520)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 92 | 70 | 46 | 145 | 31 | 101
  Change at Cycle 11 Day 1 | -2.72 (29.160) | -12.62 (27.428) | -0.36 (28.865) | 1.95 (23.032) | -12.37 (23.161) | -12.54 (26.077)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 78 | 63 | 37 | 124 | 26 | 89
  Change at Cycle 13 Day 1 | -4.27 (28.228) | -11.38 (28.053) | -0.45 (27.635) | 1.75 (24.585) | -5.77 (18.822) | -9.74 (25.723)
  Change at Cycle 15 Day 1: number analyzed (Participants) | 67 | 58 | 29 | 99 | 17 | 75
  Change at Cycle 15 Day 1 | 3.73 (25.921) | -10.63 (27.695) | -6.32 (34.622) | 2.86 (22.340) | -15.69 (16.106) | -11.78 (25.524)
  Change at Cycle 17 Day 1: number analyzed (Participants) | 60 | 54 | 24 | 63 | 14 | 68
  Change at Cycle 17 Day 1 | 1.11 (27.251) | -11.42 (25.865) | 1.39 (25.020) | 1.59 (22.543) | -7.14 (28.280) | -10.54 (26.219)
  Change at Cycle 19 Day 1: number analyzed (Participants) | 48 | 50 | 22 | 27 | 9 | 59
  Change at Cycle 19 Day 1 | -1.04 (30.248) | -12.33 (30.826) | 3.79 (26.192) | 1.23 (22.133) | -12.96 (34.134) | -12.43 (31.041)
  Change at Cycle 21 Day 1: number analyzed (Participants) | 33 | 43 | 16 | 11 | 1 | 44
  Change at Cycle 21 Day 1 | -1.52 (32.103) | -14.73 (30.257) | -3.13 (22.948) | 4.55 (18.395) | -33.33 | -15.15 (30.034)
  Change at Cycle 23 Day 1: number analyzed (Participants) | 23 | 34 | 12 | 0 | 0 | 34
  Change at Cycle 23 Day 1 | -12.32 (28.077) | -6.37 (20.521) | 1.39 (15.006) |  |  | -6.37 (20.521)
  Change at Cycle 25 Day 1: number analyzed (Participants) | 16 | 26 | 7 | 0 | 0 | 26
  Change at Cycle 25 Day 1 | -5.21 (23.348) | -7.05 (24.117) | 4.76 (20.893) |  |  | -7.05 (24.117)
  Change at End of treatment visit: number analyzed (Participants) | 2 | 7 | 4 | 4 | 3 | 10
  Change at End of treatment visit | 25.00 (35.355) | -19.05 (26.227) | -8.33 (9.623) | -16.67 (30.429) | 0.00 (33.333) | -13.33 (28.109)

32. Secondary Outcome: Part 1 and Part 2: Number of Participants With Change From Baseline in Eastern Cooperative Oncology Group Performance Status (ECOG PS)
Description: ECOG: participant's performance status was measured on a 6-point scale: 0= fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light and sedentary nature; 2= ambulatory and capable of all self-care, but unable to carry out any work activities, up and about more than 50% of waking hours; 3= capable of only limited self-care, confined to bed/chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed/chair: 5= dead.
Time Frame: Part 1 and Part 2: Baseline, Day 1 of each cycle (Cycle 2 to Cycle 31)
Population: Safety analysis set included all participants who received at least one dose of study medication and have at least one valid post-baseline safety evaluation. Here, "Number analyzed" signifies participants evaluable for each specified row. It was planned to report combined result data of Part 1 and Part 2 for LGX818 300 mg arm. Data is reported only for categories with non-zero values.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 192 | 192 | 186 | 257 | 84 | 276
Participants
  Baseline: ECOG score 0 | 136 | 139 | 135 | 189 | 60 | 199
  Baseline: ECOG score 1 | 56 | 53 | 51 | 68 | 24 | 77
  Cycle 2 Day 1: ECOG score 0: number analyzed (Participants) | 188 | 182 | 181 | 256 | 80 | 262
  Cycle 2 Day 1: ECOG score 0 | 142 | 98 | 113 | 193 | 44 | 142
  Cycle 2 Day 1: ECOG score 1: number analyzed (Participants) | 188 | 182 | 181 | 256 | 80 | 262
  Cycle 2 Day 1: ECOG score 1 | 44 | 79 | 64 | 62 | 32 | 111
  Cycle 2 Day 1: ECOG score 2: number analyzed (Participants) | 188 | 182 | 181 | 256 | 80 | 262
  Cycle 2 Day 1: ECOG score 2 | 1 | 3 | 4 | 1 | 4 | 7
  Cycle 2 Day 1: ECOG score 3: number analyzed (Participants) | 188 | 182 | 181 | 256 | 80 | 262
  Cycle 2 Day 1: ECOG score 3 | 0 | 2 | 0 | 0 | 0 | 2
  Cycle 2 Day 1: ECOG score 4: number analyzed (Participants) | 188 | 182 | 181 | 256 | 80 | 262
  Cycle 2 Day 1: ECOG score 4 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: ECOG score 0: number analyzed (Participants) | 185 | 175 | 176 | 253 | 74 | 249
  Cycle 3 Day 1: ECOG score 0 | 131 | 90 | 107 | 197 | 40 | 130
  Cycle 3 Day 1: ECOG score 1: number analyzed (Participants) | 185 | 175 | 176 | 253 | 74 | 249
  Cycle 3 Day 1: ECOG score 1 | 53 | 81 | 64 | 55 | 32 | 113
  Cycle 3 Day 1: ECOG score 2: number analyzed (Participants) | 185 | 175 | 176 | 253 | 74 | 249
  Cycle 3 Day 1: ECOG score 2 | 1 | 4 | 4 | 1 | 2 | 6
  Cycle 4 Day 1: ECOG score 0: number analyzed (Participants) | 179 | 164 | 158 | 250 | 68 | 232
  Cycle 4 Day 1: ECOG score 0 | 128 | 93 | 98 | 189 | 35 | 128
  Cycle 4 Day 1: ECOG score 1: number analyzed (Participants) | 179 | 164 | 158 | 250 | 68 | 232
  Cycle 4 Day 1: ECOG score 1 | 50 | 66 | 52 | 56 | 30 | 96
  Cycle 4 Day 1: ECOG score 2: number analyzed (Participants) | 179 | 164 | 158 | 250 | 68 | 232
  Cycle 4 Day 1: ECOG score 2 | 1 | 4 | 4 | 4 | 3 | 7
  Cycle 4 Day 1: ECOG score 3: number analyzed (Participants) | 179 | 164 | 158 | 250 | 68 | 232
  Cycle 4 Day 1: ECOG score 3 | 0 | 1 | 4 | 1 | 0 | 1
  Cycle 5 Day 1: ECOG score 0: number analyzed (Participants) | 174 | 158 | 143 | 239 | 66 | 224
  Cycle 5 Day 1: ECOG score 0 | 128 | 85 | 82 | 181 | 33 | 118
  Cycle 5 Day 1: ECOG score 1: number analyzed (Participants) | 174 | 158 | 143 | 239 | 66 | 224
  Cycle 5 Day 1: ECOG score 1 | 42 | 69 | 52 | 55 | 31 | 100
  Cycle 5 Day 1: ECOG score 2: number analyzed (Participants) | 174 | 158 | 143 | 239 | 66 | 224
  Cycle 5 Day 1: ECOG score 2 | 3 | 4 | 7 | 2 | 2 | 6
  Cycle 5 Day 1: ECOG score 3: number analyzed (Participants) | 174 | 158 | 143 | 239 | 66 | 224
  Cycle 5 Day 1: ECOG score 3 | 1 | 0 | 1 | 1 | 0 | 0
  Cycle 5 Day 1: ECOG score 4: number analyzed (Participants) | 174 | 158 | 143 | 239 | 66 | 224
  Cycle 5 Day 1: ECOG score 4 | 0 | 0 | 1 | 0 | 0 | 0
  Cycle 6 Day 1: ECOG score 0: number analyzed (Participants) | 169 | 137 | 126 | 231 | 58 | 195
  Cycle 6 Day 1: ECOG score 0 | 124 | 68 | 78 | 168 | 29 | 97
  Cycle 6 Day 1: ECOG score 1: number analyzed (Participants) | 169 | 137 | 126 | 231 | 58 | 195
  Cycle 6 Day 1: ECOG score 1 | 45 | 65 | 46 | 58 | 25 | 90
  Cycle 6 Day 1: ECOG score 2: number analyzed (Participants) | 169 | 137 | 126 | 231 | 58 | 195
  Cycle 6 Day 1: ECOG score 2 | 0 | 3 | 1 | 3 | 3 | 6
  Cycle 6 Day 1: ECOG score 3: number analyzed (Participants) | 169 | 137 | 126 | 231 | 58 | 195
  Cycle 6 Day 1: ECOG score 3 | 0 | 0 | 1 | 1 | 1 | 1
  Cycle 6 Day 1: ECOG score 4: number analyzed (Participants) | 169 | 137 | 126 | 231 | 58 | 195
  Cycle 6 Day 1: ECOG score 4 | 0 | 1 | 0 | 1 | 0 | 1
  Cycle 7 Day 1: ECOG score 0: number analyzed (Participants) | 158 | 129 | 111 | 218 | 55 | 184
  Cycle 7 Day 1: ECOG score 0 | 111 | 68 | 74 | 158 | 27 | 95
  Cycle 7 Day 1: ECOG score 1: number analyzed (Participants) | 158 | 129 | 111 | 218 | 55 | 184
  Cycle 7 Day 1: ECOG score 1 | 46 | 60 | 35 | 58 | 27 | 87
  Cycle 7 Day 1: ECOG score 2: number analyzed (Participants) | 158 | 129 | 111 | 218 | 55 | 184
  Cycle 7 Day 1: ECOG score 2 | 1 | 1 | 2 | 2 | 1 | 2
  Cycle 8 Day 1: ECOG score 0: number analyzed (Participants) | 148 | 108 | 95 | 200 | 46 | 154
  Cycle 8 Day 1: ECOG score 0 | 112 | 55 | 58 | 140 | 22 | 77
  Cycle 8 Day 1: ECOG score 1: number analyzed (Participants) | 148 | 108 | 95 | 200 | 46 | 154
  Cycle 8 Day 1: ECOG score 1 | 33 | 49 | 33 | 58 | 21 | 70
  Cycle 8 Day 1: ECOG score 2: number analyzed (Participants) | 148 | 108 | 95 | 200 | 46 | 154
  Cycle 8 Day 1: ECOG score 2 | 2 | 3 | 4 | 1 | 3 | 6
  Cycle 8 Day 1: ECOG score 3: number analyzed (Participants) | 148 | 108 | 95 | 200 | 46 | 154
  Cycle 8 Day 1: ECOG score 3 | 1 | 1 | 0 | 1 | 0 | 1
  Cycle 9 Day 1: ECOG score 0: number analyzed (Participants) | 144 | 98 | 90 | 188 | 43 | 141
  Cycle 9 Day 1: ECOG score 0 | 102 | 50 | 55 | 135 | 22 | 72
  Cycle 9 Day 1: ECOG score 1: number analyzed (Participants) | 144 | 98 | 90 | 188 | 43 | 141
  Cycle 9 Day 1: ECOG score 1 | 36 | 47 | 30 | 52 | 20 | 67
  Cycle 9 Day 1: ECOG score 2: number analyzed (Participants) | 144 | 98 | 90 | 188 | 43 | 141
  Cycle 9 Day 1: ECOG score 2 | 4 | 1 | 4 | 0 | 0 | 1
  Cycle 9 Day 1: ECOG score 3: number analyzed (Participants) | 144 | 98 | 90 | 188 | 43 | 141
  Cycle 9 Day 1: ECOG score 3 | 0 | 0 | 1 | 0 | 1 | 1
  Cycle 9 Day 1: ECOG score 4: number analyzed (Participants) | 144 | 98 | 90 | 188 | 43 | 141
  Cycle 9 Day 1: ECOG score 4 | 1 | 0 | 0 | 1 | 0 | 0
  Cycle 9 Day 1: ECOG score 5: number analyzed (Participants) | 144 | 98 | 90 | 188 | 43 | 141
  Cycle 9 Day 1: ECOG score 5 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: ECOG score 0: number analyzed (Participants) | 129 | 88 | 72 | 171 | 37 | 125
  Cycle 10 Day 1: ECOG score 0 | 94 | 52 | 43 | 121 | 18 | 70
  Cycle 10 Day 1: ECOG score 1: number analyzed (Participants) | 129 | 88 | 72 | 171 | 37 | 125
  Cycle 10 Day 1: ECOG score 1 | 32 | 35 | 26 | 46 | 18 | 53
  Cycle 10 Day 1: ECOG score 2: number analyzed (Participants) | 129 | 88 | 72 | 171 | 37 | 125
  Cycle 10 Day 1: ECOG score 2 | 3 | 1 | 2 | 3 | 1 | 2
  Cycle 10 Day 1: ECOG score 3: number analyzed (Participants) | 129 | 88 | 72 | 171 | 37 | 125
  Cycle 10 Day 1: ECOG score 3 | 0 | 0 | 1 | 1 | 0 | 0
  Cycle 11 Day 1: ECOG score 0: number analyzed (Participants) | 120 | 85 | 62 | 158 | 36 | 121
  Cycle 11 Day 1: ECOG score 0 | 88 | 44 | 39 | 116 | 17 | 61
  Cycle 11 Day 1: ECOG score 1: number analyzed (Participants) | 120 | 85 | 62 | 158 | 36 | 121
  Cycle 11 Day 1: ECOG score 1 | 30 | 40 | 20 | 42 | 16 | 56
  Cycle 11 Day 1: ECOG score 2: number analyzed (Participants) | 120 | 85 | 62 | 158 | 36 | 121
  Cycle 11 Day 1: ECOG score 2 | 2 | 1 | 2 | 0 | 3 | 4
  Cycle 11 Day 1: ECOG score 3: number analyzed (Participants) | 120 | 85 | 62 | 158 | 36 | 121
  Cycle 11 Day 1: ECOG score 3 | 0 | 0 | 1 | 0 | 0 | 0
  Cycle 12 Day 1: ECOG score 0: number analyzed (Participants) | 110 | 77 | 51 | 152 | 30 | 107
  Cycle 12 Day 1: ECOG score 0 | 84 | 44 | 32 | 113 | 11 | 55
  Cycle 12 Day 1: ECOG score 1: number analyzed (Participants) | 110 | 77 | 51 | 152 | 30 | 107
  Cycle 12 Day 1: ECOG score 1 | 25 | 31 | 16 | 38 | 18 | 49
  Cycle 12 Day 1: ECOG score 2: number analyzed (Participants) | 110 | 77 | 51 | 152 | 30 | 107
  Cycle 12 Day 1: ECOG score 2 | 1 | 1 | 2 | 0 | 1 | 2
  Cycle 12 Day 1: ECOG score 3: number analyzed (Participants) | 110 | 77 | 51 | 152 | 30 | 107
  Cycle 12 Day 1: ECOG score 3 | 0 | 1 | 1 | 0 | 0 | 1
  Cycle 12 Day 1: ECOG score 4: number analyzed (Participants) | 110 | 77 | 51 | 152 | 30 | 107
  Cycle 12 Day 1: ECOG score 4 | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 13 Day 1: ECOG score 0: number analyzed (Participants) | 100 | 73 | 47 | 143 | 31 | 104
  Cycle 13 Day 1: ECOG score 0 | 77 | 41 | 27 | 102 | 14 | 55
  Cycle 13 Day 1: ECOG score 1: number analyzed (Participants) | 100 | 73 | 47 | 143 | 31 | 104
  Cycle 13 Day 1: ECOG score 1 | 22 | 31 | 18 | 39 | 15 | 46
  Cycle 13 Day 1: ECOG score 2: number analyzed (Participants) | 100 | 73 | 47 | 143 | 31 | 104
  Cycle 13 Day 1: ECOG score 2 | 1 | 1 | 2 | 1 | 2 | 3
  Cycle 13 Day 1: ECOG score 4: number analyzed (Participants) | 100 | 73 | 47 | 143 | 31 | 104
  Cycle 13 Day 1: ECOG score 4 | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 14 Day 1: ECOG score 0: number analyzed (Participants) | 97 | 75 | 46 | 136 | 27 | 102
  Cycle 14 Day 1: ECOG score 0 | 74 | 47 | 25 | 100 | 15 | 62
  Cycle 14 Day 1: ECOG score 1: number analyzed (Participants) | 97 | 75 | 46 | 136 | 27 | 102
  Cycle 14 Day 1: ECOG score 1 | 23 | 27 | 19 | 33 | 10 | 37
  Cycle 14 Day 1: ECOG score 2: number analyzed (Participants) | 97 | 75 | 46 | 136 | 27 | 102
  Cycle 14 Day 1: ECOG score 2 | 0 | 0 | 2 | 2 | 2 | 2
  Cycle 14 Day 1: ECOG score 3: number analyzed (Participants) | 97 | 75 | 46 | 136 | 27 | 102
  Cycle 14 Day 1: ECOG score 3 | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 14 Day 1: ECOG score 4: number analyzed (Participants) | 97 | 75 | 46 | 136 | 27 | 102
  Cycle 14 Day 1: ECOG score 4 | 0 | 1 | 0 | 0 | 0 | 1
  Cycle 15 Day 1: ECOG score 0: number analyzed (Participants) | 94 | 72 | 41 | 111 | 21 | 93
  Cycle 15 Day 1: ECOG score 0 | 72 | 41 | 22 | 82 | 13 | 54
  Cycle 15 Day 1: ECOG score 1: number analyzed (Participants) | 94 | 72 | 41 | 111 | 21 | 93
  Cycle 15 Day 1: ECOG score 1 | 20 | 30 | 18 | 27 | 7 | 37
  Cycle 15 Day 1: ECOG score 2: number analyzed (Participants) | 94 | 72 | 41 | 111 | 21 | 93
  Cycle 15 Day 1: ECOG score 2 | 1 | 1 | 1 | 1 | 1 | 2
  Cycle 15 Day 1: ECOG score 3: number analyzed (Participants) | 94 | 72 | 41 | 111 | 21 | 93
  Cycle 15 Day 1: ECOG score 3 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 15 Day 1: ECOG score 4: number analyzed (Participants) | 94 | 72 | 41 | 111 | 21 | 93
  Cycle 15 Day 1: ECOG score 4 | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 16 Day 1: ECOG score 0: number analyzed (Participants) | 89 | 67 | 35 | 88 | 19 | 86
  Cycle 16 Day 1: ECOG score 0 | 64 | 41 | 24 | 64 | 11 | 52
  Cycle 16 Day 1: ECOG score 1: number analyzed (Participants) | 89 | 67 | 35 | 88 | 19 | 86
  Cycle 16 Day 1: ECOG score 1 | 24 | 23 | 10 | 23 | 7 | 30
  Cycle 16 Day 1: ECOG score 2: number analyzed (Participants) | 89 | 67 | 35 | 88 | 19 | 86
  Cycle 16 Day 1: ECOG score 2 | 1 | 3 | 1 | 0 | 1 | 4
  Cycle 16 Day 1: ECOG score 3: number analyzed (Participants) | 89 | 67 | 35 | 88 | 19 | 86
  Cycle 16 Day 1: ECOG score 3 | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 17 Day 1: ECOG score 0: number analyzed (Participants) | 82 | 67 | 33 | 68 | 16 | 83
  Cycle 17 Day 1: ECOG score 0 | 65 | 39 | 21 | 52 | 9 | 48
  Cycle 17 Day 1: ECOG score 1: number analyzed (Participants) | 82 | 67 | 33 | 68 | 16 | 83
  Cycle 17 Day 1: ECOG score 1 | 16 | 27 | 11 | 15 | 6 | 33
  Cycle 17 Day 1: ECOG score 2: number analyzed (Participants) | 82 | 67 | 33 | 68 | 16 | 83
  Cycle 17 Day 1: ECOG score 2 | 1 | 1 | 1 | 1 | 1 | 2
  Cycle 18 Day 1: ECOG score 0: number analyzed (Participants) | 75 | 60 | 31 | 46 | 10 | 70
  Cycle 18 Day 1: ECOG score 0 | 60 | 36 | 18 | 34 | 5 | 41
  Cycle 18 Day 1: ECOG score 1: number analyzed (Participants) | 75 | 60 | 31 | 46 | 10 | 70
  Cycle 18 Day 1: ECOG score 1 | 14 | 24 | 11 | 11 | 5 | 29
  Cycle 18 Day 1: ECOG score 2: number analyzed (Participants) | 75 | 60 | 31 | 46 | 10 | 70
  Cycle 18 Day 1: ECOG score 2 | 1 | 0 | 1 | 1 | 0 | 0
  Cycle 18 Day 1: ECOG score 3: number analyzed (Participants) | 75 | 60 | 31 | 46 | 10 | 70
  Cycle 18 Day 1: ECOG score 3 | 0 | 0 | 1 | 0 | 0 | 0
  Cycle 19 Day 1: ECOG score 0: number analyzed (Participants) | 65 | 59 | 30 | 30 | 8 | 67
  Cycle 19 Day 1: ECOG score 0 | 54 | 38 | 20 | 22 | 2 | 40
  Cycle 19 Day 1: ECOG score 1: number analyzed (Participants) | 65 | 59 | 30 | 30 | 8 | 67
  Cycle 19 Day 1: ECOG score 1 | 9 | 20 | 9 | 7 | 6 | 26
  Cycle 19 Day 1: ECOG score 2: number analyzed (Participants) | 65 | 59 | 30 | 30 | 8 | 67
  Cycle 19 Day 1: ECOG score 2 | 2 | 1 | 1 | 1 | 0 | 1
  Cycle 20 Day 1: ECOG score 0: number analyzed (Participants) | 61 | 52 | 27 | 20 | 6 | 58
  Cycle 20 Day 1: ECOG score 0 | 53 | 31 | 19 | 15 | 3 | 34
  Cycle 20 Day 1: ECOG score 1: number analyzed (Participants) | 61 | 52 | 27 | 20 | 6 | 58
  Cycle 20 Day 1: ECOG score 1 | 7 | 19 | 8 | 5 | 3 | 22
  Cycle 20 Day 1: ECOG score 2: number analyzed (Participants) | 61 | 52 | 27 | 20 | 6 | 58
  Cycle 20 Day 1: ECOG score 2 | 0 | 2 | 0 | 0 | 0 | 2
  Cycle 20 Day 1: ECOG score 3: number analyzed (Participants) | 61 | 52 | 27 | 20 | 6 | 58
  Cycle 20 Day 1: ECOG score 3 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 21 Day 1: ECOG score 0: number analyzed (Participants) | 46 | 49 | 23 | 13 | 3 | 52
  Cycle 21 Day 1: ECOG score 0 | 36 | 29 | 15 | 11 | 2 | 31
  Cycle 21 Day 1: ECOG score 1: number analyzed (Participants) | 46 | 49 | 23 | 13 | 3 | 52
  Cycle 21 Day 1: ECOG score 1 | 10 | 19 | 8 | 2 | 1 | 20
  Cycle 21 Day 1: ECOG score 2: number analyzed (Participants) | 46 | 49 | 23 | 13 | 3 | 52
  Cycle 21 Day 1: ECOG score 2 | 9 | 1 | 0 | 0 | 0 | 1
  Cycle 22 Day 1: ECOG score 0: number analyzed (Participants) | 37 | 45 | 17 | 6 | 0 | 45
  Cycle 22 Day 1: ECOG score 0 | 29 | 27 | 11 | 4 | 0 | 27
  Cycle 22 Day 1: ECOG score 1: number analyzed (Participants) | 37 | 45 | 17 | 6 | 0 | 45
  Cycle 22 Day 1: ECOG score 1 | 8 | 16 | 6 | 2 | 0 | 16
  Cycle 22 Day 1: ECOG score 3: number analyzed (Participants) | 37 | 45 | 17 | 6 | 0 | 45
  Cycle 22 Day 1: ECOG score 3 | 0 | 1 | 0 | 0 | 0 | 1
  Cycle 22 Day 1: ECOG score 4: number analyzed (Participants) | 37 | 45 | 17 | 6 | 0 | 45
  Cycle 22 Day 1: ECOG score 4 | 0 | 1 | 0 | 0 | 0 | 1
  Cycle 23 Day 1: ECOG score 0: number analyzed (Participants) | 30 | 38 | 15 | 0 | 0 | 38
  Cycle 23 Day 1: ECOG score 0 | 24 | 26 | 10 | 0 | 0 | 26
  Cycle 23 Day 1: ECOG score 1: number analyzed (Participants) | 30 | 38 | 15 | 0 | 0 | 38
  Cycle 23 Day 1: ECOG score 1 | 6 | 12 | 5 | 0 | 0 | 12
  Cycle 24 Day 1: ECOG score 0: number analyzed (Participants) | 28 | 33 | 14 | 0 | 0 | 33
  Cycle 24 Day 1: ECOG score 0 | 21 | 23 | 9 | 0 | 0 | 23
  Cycle 24 Day 1: ECOG score 1: number analyzed (Participants) | 28 | 33 | 14 | 0 | 0 | 33
  Cycle 24 Day 1: ECOG score 1 | 7 | 10 | 5 | 0 | 0 | 10
  Cycle 25 Day 1: ECOG score 0: number analyzed (Participants) | 20 | 31 | 11 | 0 | 0 | 31
  Cycle 25 Day 1: ECOG score 0 | 17 | 23 | 9 | 0 | 0 | 23
  Cycle 25 Day 1: ECOG score 1: number analyzed (Participants) | 20 | 31 | 11 | 0 | 0 | 31
  Cycle 25 Day 1: ECOG score 1 | 3 | 8 | 2 | 0 | 0 | 8
  Cycle 26 Day 1: ECOG score 0: number analyzed (Participants) | 18 | 29 | 9 | 0 | 0 | 29
  Cycle 26 Day 1: ECOG score 0 | 14 | 21 | 7 | 0 | 0 | 21
  Cycle 26 Day 1: ECOG score 1: number analyzed (Participants) | 18 | 29 | 9 | 0 | 0 | 29
  Cycle 26 Day 1: ECOG score 1 | 3 | 8 | 2 | 0 | 0 | 8
  Cycle 26 Day 1: ECOG score 2: number analyzed (Participants) | 18 | 29 | 9 | 0 | 0 | 29
  Cycle 26 Day 1: ECOG score 2 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 27 Day 1: ECOG score 0: number analyzed (Participants) | 8 | 26 | 7 | 0 | 0 | 26
  Cycle 27 Day 1: ECOG score 0 | 5 | 20 | 3 | 0 | 0 | 20
  Cycle 27 Day 1: ECOG score 1: number analyzed (Participants) | 8 | 26 | 7 | 0 | 0 | 26
  Cycle 27 Day 1: ECOG score 1 | 3 | 6 | 4 | 0 | 0 | 6
  Cycle 28 Day 1: ECOG score 0: number analyzed (Participants) | 8 | 24 | 5 | 0 | 0 | 24
  Cycle 28 Day 1: ECOG score 0 | 5 | 18 | 4 | 0 | 0 | 18
  Cycle 28 Day 1: ECOG score 1: number analyzed (Participants) | 8 | 24 | 5 | 0 | 0 | 24
  Cycle 28 Day 1: ECOG score 1 | 3 | 6 | 1 | 0 | 0 | 6
  Cycle 29 Day 1: ECOG score 0: number analyzed (Participants) | 3 | 18 | 5 | 0 | 0 | 18
  Cycle 29 Day 1: ECOG score 0 | 1 | 13 | 5 | 0 | 0 | 13
  Cycle 29 Day 1: ECOG score 1: number analyzed (Participants) | 3 | 18 | 5 | 0 | 0 | 18
  Cycle 29 Day 1: ECOG score 1 | 2 | 5 | 0 | 0 | 0 | 5
  Cycle 30 Day 1: ECOG score 0: number analyzed (Participants) | 0 | 12 | 4 | 0 | 0 | 12
  Cycle 30 Day 1: ECOG score 0 | 0 | 9 | 4 | 0 | 0 | 9
  Cycle 30 Day 1: ECOG score 1: number analyzed (Participants) | 0 | 12 | 4 | 0 | 0 | 12
  Cycle 30 Day 1: ECOG score 1 | 0 | 3 | 0 | 0 | 0 | 3
  Cycle 31 Day 1: ECOG score 0: number analyzed (Participants) | 0 | 10 | 2 | 0 | 0 | 10
  Cycle 31 Day 1: ECOG score 0 | 0 | 7 | 2 | 0 | 0 | 7
  Cycle 31 Day 1: ECOG score 1: number analyzed (Participants) | 0 | 10 | 2 | 0 | 0 | 10
  Cycle 31 Day 1: ECOG score 1 | 0 | 3 | 0 | 0 | 0 | 3

33. Secondary Outcome: Part 1: Plasma Concentrations of LGX 818
Time Frame: Cycle 1 Day 1: pre-dose, 0.5, 1.5, 4 to 8 hours post dose; Cycle 2 Day 1: pre-dose; Cycle 3 Day 1: pre-dose
Population: Pharmacokinetic analysis set included all participants who received at least one dose of LGX818 or MEK162 and had at least one evaluable post-baseline LGX818 or MEK162 concentration measurement. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number analyzed" signifies participants evaluable for each specified category at each specified row.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg
Number analyzed (Participants) | 175 | 172
nanogram per milliliter
  Cycle 1 Day 1: pre-dose | 18.6 (125) | 58.1 (513)
  Cycle 1 Day 1: 0.5 hours post dose: number analyzed (Participants) | 159 | 145
  Cycle 1 Day 1: 0.5 hours post dose | 1640 (2400) | 1190 (1790)
  Cycle 1 Day 1: 1.5 hours post dose: number analyzed (Participants) | 122 | 116
  Cycle 1 Day 1: 1.5 hours post dose | 6860 (3680) | 4090 (2100)
  Cycle 1 Day 1: 4 to 8 hours post dose: number analyzed (Participants) | 147 | 142
  Cycle 1 Day 1: 4 to 8 hours post dose | 3400 (2010) | 1850 (925)
  Cycle 2 Day 1: pre-dose: number analyzed (Participants) | 119 | 73
  Cycle 2 Day 1: pre-dose | 119 (468) | 73.6 (405)
  Cycle 3 Day 1: pre-dose: number analyzed (Participants) | 98 | 74
  Cycle 3 Day 1: pre-dose | 150 (697) | 53.8 (256)

34. Secondary Outcome: Part 2: Plasma Concentrations of LGX 818
Time Frame: Cycle 1 Day 1: pre-dose, 0.5, 1.5, 4 to 8 hours post dose; Cycle 2 Day 1: pre-dose; Cycle 3 Day 1: pre-dose
Population: Pharmacokinetic analysis set included all participants who received at least one dose of LGX818 or MEK162 and had at least one evaluable post-baseline LGX818 or MEK162 concentration measurement. Here, "Overall Number of Participants Analyzed" =number of participants evaluable for this outcome measure and "Number analyzed" =participants evaluable at each specified row. It was planned to report combined result data of Part 1 and Part 2 for LGX818 300 mg arm.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 242 | 80 | 252
nanogram per milliliter
  Cycle 1 Day 1: pre-dose | 5.02 (77.8) | 0.0145 (0.130) | 39.7 (424)
  Cycle 1 Day 1: 0.5 hours post dose: number analyzed (Participants) | 207 | 68 | 213
  Cycle 1 Day 1: 0.5 hours post dose | 1360 (2000) | 1370 (2170) | 1250 (1910)
  Cycle 1 Day 1: 1.5 hours post dose: number analyzed (Participants) | 220 | 73 | 189
  Cycle 1 Day 1: 1.5 hours post dose | 4390 (2380) | 4310 (2570) | 4170 (2290)
  Cycle 1 Day 1: 4 to 8 hours post dose: number analyzed (Participants) | 185 | 66 | 208
  Cycle 1 Day 1: 4 to 8 hours post dose | 2420 (1270) | 2250 (1170) | 1980 (1020)
  Cycle 2 Day 1: pre-dose: number analyzed (Participants) | 175 | 32 | 105
  Cycle 2 Day 1: pre-dose | 121 (483) | 29.5 (99.9) | 60.1 (342)
  Cycle 3 Day 1: pre-dose: number analyzed (Participants) | 151 | 27 | 101
  Cycle 3 Day 1: pre-dose | 74.1 (322) | 79.5 (291) | 60.6 (265)

35. Secondary Outcome: Part 1: Plasma Concentrations of MEK162
Time Frame: Cycle 1 Day 1: pre-dose, 0.5, 1.5, 4 to 8, hours post dose; Cycle 2 Day 1: pre-dose; Cycle 3 Day 1: pre-dose
Population: Pharmacokinetic analysis set included all participants who received at least one dose of LGX818 or MEK162 and had at least one evaluable post-baseline LGX818 or MEK162 concentration measurement. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number analyzed" signifies participants evaluable for each specified row.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450)
Number analyzed (Participants) | 167
nanogram per milliliter
  Cycle 1 Day 1: pre-dose | 2.95 (30.7)
  Cycle 1 Day 1: 0.5 hours post dose: number analyzed (Participants) | 151
  Cycle 1 Day 1: 0.5 hours post dose | 426 (410)
  Cycle 1 Day 1: 1.5 hours post dose: number analyzed (Participants) | 117
  Cycle 1 Day 1: 1.5 hours post dose | 832 (527)
  Cycle 1 Day 1: 4 to 8 hours post dose: number analyzed (Participants) | 138
  Cycle 1 Day 1: 4 to 8 hours post dose | 330 (226)
  Cycle 2 Day 1: pre-dose: number analyzed (Participants) | 77
  Cycle 2 Day 1: pre-dose | 81.0 (106)
  Cycle 3 Day 1: pre-dose: number analyzed (Participants) | 65
  Cycle 3 Day 1: pre-dose | 68.1 (101)

36. Secondary Outcome: Part 2: Plasma Concentrations of MEK162
Time Frame: Cycle 1 Day 1: pre-dose, 0.5, 1.5, 4 to 8, hours post dose; Cycle 2 Day 1: pre-dose; Cycle 3 Day 1: pre-dose
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300)
Number analyzed (Participants) | 215
nanogram per milliliter
  Cycle 1 Day 1: pre-dose | 1.68 (24.3)
  Cycle 1 Day 1: 0.5 hours post dose: number analyzed (Participants) | 191
  Cycle 1 Day 1: 0.5 hours post dose | 366 (347)
  Cycle 1 Day 1: 1.5 hours post dose: number analyzed (Participants) | 196
  Cycle 1 Day 1: 1.5 hours post dose | 642 (337)
  Cycle 1 Day 1: 4 to 8 hours post dose: number analyzed (Participants) | 169
  Cycle 1 Day 1: 4 to 8 hours post dose | 287 (175)
  Cycle 2 Day 1: pre-dose: number analyzed (Participants) | 98
  Cycle 2 Day 1: pre-dose | 72.3 (62.6)
  Cycle 3 Day 1: pre-dose: number analyzed (Participants) | 94
  Cycle 3 Day 1: pre-dose | 73.2 (89.0)

37. Secondary Outcome: Part 1 and Part 2: Time to Definitive 1 Point Deterioration in Eastern Cooperative Oncology Group Performance Status (ECOG PS)
Description: ECOG: participant's performance status was measured on a 6-point scale: 0= fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light and sedentary nature; 2= ambulatory and capable of all self-care, but unable to carry out any work activities, up and about more than 50 percent (%) of waking hours; 3= capable of only limited self-care, confined to bed/chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed/chair: 5= dead. Definitive deterioration was defined as death due to any cause or decrease in ECOG PS by at least one category from baseline score with no subsequent improvement.
Time Frame: Baseline up to 30 days from last dose of study drug (up to 30 months for Part 1, excluding Part 1: LGX818 300 mg group; up to 36 months for Part 2 and Part 1 LGX 300 mg group)
Population: Safety analysis set includes all participants who received at least one dose of study medication and have at least one valid post-baseline safety evaluation. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. It was planned to report combined result data of Part 1 and Part 2 for LGX818 300 mg arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1:LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg | Part 1 + Part 2: LGX818 300 mg
Number analyzed (Participants) | 192 | 187 | 185 | 257 | 83 | 270
months | NA [23.0 to NA] — Median and upper limit of 95% CI were not estimable due to low number of participants with events. | 26.7 [14.8 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | 18.2 [11.1 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | NA [NA to NA] — Median and 95% CI were not estimable due to low number of participants with events. | 10.2 [8.1 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | 19.2 [12.9 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events.

ADVERSE EVENTS:
Time Frame: Part 1: Baseline up to 30 days from last dose of study drug (up to 30 months for Part 1, excluding Part 1: LGX818 300 mg group; up to 36 months for Part 2 and Part 1 LGX 300 mg group)
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis population evaluated.
Arm/Group | Part 1: LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) | Part 1: LGX818 300 mg | Part 1: Vemurafenib 960 mg BID | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) | Part 2: LGX818 300 mg
Serious Adverse Events (participants affected / at risk) | 66/192 | 67/192 | 69/186 | 75/257 | 25/84
Other Adverse Events (participants affected / at risk) | 189/192 | 190/192 | 184/186 | 251/257 | 81/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) (N=192) | Part 1: LGX818 300 mg (N=192) | Part 1: Vemurafenib 960 mg BID (N=186) | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) (N=257) | Part 2: LGX818 300 mg (N=84)
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 2 | 4 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 0 | 0 | 3 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 0 | 1 | 0
Atrioventricular Block First Degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Bundle Branch Block Left (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Left Ventricular Failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Chorioretinopathy (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal Detachment (Eye disorders) | 1 | 0 | 0 | 1 | 0
Normal Tension Glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 0
Retinal Artery Occlusion (Eye disorders) | 0 | 1 | 0 | 0 | 0
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 4 | 2 | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 3 | 6 | 2 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 6 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anal Incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 6 | 3 | 2 | 2 | 0
General Physical Health Deterioration (General disorders) | 3 | 2 | 6 | 4 | 1
Death (General disorders) | 2 | 1 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 2 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 4 | 0 | 1 | 0
Gait Disturbance (General disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Contrast Media Allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 2 | 0
Erysipelas (Infections and infestations) | 2 | 1 | 0 | 3 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 0 | 1 | 0
Campylobacter Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis Streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Chorioretinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Escherichia Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infected Seroma (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Intestinal Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Peritonsillar Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Streptococcal Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radiation Necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Blood Creatinine Increased (Investigations) | 1 | 0 | 0 | 1 | 0
C-Reactive Protein Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 1 | 1 | 1 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Intraocular Pressure Increased (Investigations) | 0 | 1 | 0 | 0 | 0
Lipase Increased (Investigations) | 0 | 1 | 0 | 0 | 0
Lymph Node Palpable (Investigations) | 0 | 0 | 1 | 0 | 0
Myocardial Necrosis Marker Increased (Investigations) | 0 | 1 | 0 | 0 | 0
White Blood Cell Count Increased (Investigations) | 0 | 0 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 1 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Fracture Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1 | 1
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Intracranial Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 2 | 3 | 1
Metastases To Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 0
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Dermatofibrosarcoma Protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0
Malignant Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Metastases To Adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Superficial Spreading Melanoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 3 | 2 | 1 | 0 | 1
Balance Disorder (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Cervicobrachial Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Coma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 1 | 2 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 2 | 3 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 2 | 0
Brain Oedema (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Brain Stem Syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Facial Paralysis (Nervous system disorders) | 0 | 3 | 0 | 0 | 1
Facial Paresis (Nervous system disorders) | 0 | 2 | 0 | 0 | 2
Glial Scar (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Intercostal Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Intracranial Pressure Increased (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nervous System Disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Restless Legs Syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 1 | 4 | 0
Device Failure (Product Issues) | 0 | 1 | 0 | 0 | 0
Completed Suicide (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression Suicidal (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 3 | 1 | 1 | 2 | 3
Calculus Urethral (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 1 | 2 | 1 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary Tract Disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Ureteric Obstruction (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Breast Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 0 | 0
Mediastinal Shift (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary Alveolar Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0
Cutaneous Vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Granuloma Annulare (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash Generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Thrombophlebitis Superficial (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac Tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 0 | 3 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1 | 0
Retinal Vein Occlusion (Eye disorders) | 0 | 0 | 0 | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Performance Status Decreased (General disorders) | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Flavivirus Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Liver Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Myelitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Peritoneal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Acetabulum Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Anticoagulation Drug Level Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Troponin Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Metastases To Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Metastases To Spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebellar Ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Depressed Level Of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Facial Nerve Disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Guillain-Barre Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypertensive Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paresis Cranial Nerve (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Speech Disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Vertebral Artery Dissection (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Diplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Monoplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Post-Traumatic Stress Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Circulatory Collapse (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Motor Dysfunction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: LGX818 450 mg QD+MEK162 45 mg BID (Combo 450) (N=192) | Part 1: LGX818 300 mg (N=192) | Part 1: Vemurafenib 960 mg BID (N=186) | Part 2: LGX818 300 mg QD+MEK162 45 mg BID (Combo 300) (N=257) | Part 2: LGX818 300 mg (N=84)
Anaemia (Blood and lymphatic system disorders) | 29 | 11 | 14 | 23 | 5
Vision blurred (Eye disorders) | 30 | 4 | 4 | 26 | 2
Retinal detachment (Eye disorders) | 15 | 1 | 1 | 19 | 0
Cataract (Eye disorders) | 12 | 2 | 4 | 0 | 0
Dry eye (Eye disorders) | 11 | 10 | 12 | 0 | 0
Macular oedema (Eye disorders) | 11 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 78 | 69 | 63 | 68 | 24
Diarrhoea (Gastrointestinal disorders) | 69 | 26 | 63 | 73 | 6
Vomiting (Gastrointestinal disorders) | 57 | 47 | 27 | 39 | 16
Constipation (Gastrointestinal disorders) | 42 | 27 | 12 | 43 | 9
Abdominal pain (Gastrointestinal disorders) | 30 | 11 | 11 | 26 | 5
Abdominal pain upper (Gastrointestinal disorders) | 21 | 16 | 17 | 32 | 4
Dyspepsia (Gastrointestinal disorders) | 11 | 7 | 8 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 15 | 11 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 7 | 10 | 0 | 0
Fatigue (General disorders) | 54 | 48 | 56 | 57 | 25
Asthenia (General disorders) | 35 | 36 | 34 | 38 | 13
Pyrexia (General disorders) | 31 | 27 | 51 | 43 | 11
Oedema peripheral (General disorders) | 20 | 15 | 20 | 28 | 3
Chills (General disorders) | 9 | 11 | 10 | 0 | 0
Influenza like illness (General disorders) | 9 | 10 | 3 | 0 | 0
Xerosis (General disorders) | 4 | 16 | 8 | 0 | 0
Nasopharyngitis (Infections and infestations) | 20 | 11 | 18 | 23 | 5
Upper respiratory tract infection (Infections and infestations) | 14 | 5 | 5 | 0 | 0
Influenza (Infections and infestations) | 10 | 6 | 8 | 0 | 0
Folliculitis (Infections and infestations) | 5 | 8 | 10 | 0 | 0
Conjunctivitis (Infections and infestations) | 4 | 8 | 14 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 19 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 44 | 2 | 4 | 51 | 0
Gamma-glutamyltransferase increased (Investigations) | 29 | 20 | 20 | 36 | 7
Alanine aminotransferase increased (Investigations) | 21 | 10 | 14 | 29 | 1
Aspartate aminotransferase increased (Investigations) | 16 | 8 | 15 | 21 | 1
Blood alkaline phosphatase increased (Investigations) | 16 | 6 | 9 | 0 | 0
Blood creatinine increased (Investigations) | 11 | 3 | 11 | 0 | 0
Ejection fraction decreased (Investigations) | 11 | 4 | 1 | 0 | 0
Weight decreased (Investigations) | 6 | 29 | 20 | 10 | 8
Blood bilirubin increased (Investigations) | 2 | 0 | 14 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 16 | 40 | 36 | 23 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 49 | 84 | 81 | 57 | 35
Myalgia (Musculoskeletal and connective tissue disorders) | 26 | 53 | 34 | 35 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 41 | 24 | 27 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 26 | 10 | 36 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 6 | 4 | 18 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 30 | 10 | 9 | 10
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 18 | 31 | 16 | 13
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 12 | 10 | 6 | 5
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 12 | 21 | 4 | 10
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 18 | 7 | 4 | 5
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 10 | 0 | 0
Headache (Nervous system disorders) | 41 | 51 | 35 | 30 | 19
Dizziness (Nervous system disorders) | 23 | 9 | 5 | 21 | 1
Visual field defect (Nervous system disorders) | 14 | 2 | 3 | 0 | 0
Paraesthesia (Nervous system disorders) | 11 | 14 | 10 | 7 | 7
Dysgeusia (Nervous system disorders) | 10 | 22 | 16 | 9 | 5
Insomnia (Psychiatric disorders) | 18 | 35 | 15 | 17 | 12
Anxiety (Psychiatric disorders) | 12 | 7 | 4 | 5 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 17 | 12 | 15 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 8 | 14 | 10 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 9 | 12 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 27 | 58 | 42 | 21 | 19
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 27 | 72 | 54 | 25 | 35
Rash (Skin and subcutaneous tissue disorders) | 27 | 41 | 54 | 18 | 23
Alopecia (Skin and subcutaneous tissue disorders) | 26 | 107 | 68 | 33 | 28
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 42 | 20 | 19 | 10
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 17 | 49 | 29 | 17 | 16
Erythema (Skin and subcutaneous tissue disorders) | 13 | 24 | 31 | 14 | 11
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13 | 98 | 26 | 10 | 31
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 9 | 33 | 43 | 5 | 10
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 8 | 7 | 45 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 5 | 4 | 10 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4 | 18 | 19 | 6 | 9
Rash generalised (Skin and subcutaneous tissue disorders) | 4 | 12 | 16 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 18 | 27 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 | 15 | 3 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 10 | 6 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 9 | 12 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 11 | 4 | 0 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 15 | 0 | 0
Hypertension (Vascular disorders) | 21 | 11 | 21 | 20 | 4
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 5
Pain (General disorders) | 0 | 0 | 0 | 5 | 7
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 13 | 3
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 5 | 5
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 5
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.